

Title: A Single-Sequence, Open-Label, 2-Period, Crossover Study to Evaluate the Effect of the Proton Pump Inhibitor Esomeprazole on the Single-Dose Pharmacokinetics of Oral TAK-906 in Healthy Adult Subjects

NCT Number: NCT03849690

Protocol Approve Date: 4 Feb 2019

Certain information within this protocol has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information (PPD) or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

PROTOCOL

Single-Sequence, Open-Label, 2-Period, Crossover Study to Evaluate the Effect of the Proton Pump Inhibitor Esomeprazole on the Single-Dose Pharmacokinetics of Oral TAK-906 in Healthy Adult Subjects et of takeda. For noncommercial use only and subject to the adopticable property of takeda. For noncommercial use A Single-Sequence, Open-Label, 2-Period, Crossover Study to Evaluate the Effect of the

## **TABLE OF CONTENTS**

| 1.0 | STUDY SUMMARY | 6 |
|---|---|---|
| 2.0 | STUDY SCHEMATIC | 10 |
| 3.0 | SCHEDULE OF STUDY PROCEDURES | 12 |
| 4.0 | INTRODUCTION | 14 |
| 4. | 1 Background for TAK-906 | 14 |
| 4. | 2 Background for Esomeprazole | 14 |
| 4 | Rationale for the Proposed Study | 15 |
| 4.4 | | 15 |
| 5.0 | STUDY OBJECTIVES AND ENDPOINTS | 17 |
| 5. | 1 Hypothesis | 17 |
| 5 | 2 Study Objectives | 17 |
| | 5.2.1 Study Primary Objective | 17 |
| | STUDY OBJECTIVES AND ENDPOINTS 1 Hypothesis 2 Study Objectives 5.2.1 Study Primary Objective 5.2.2 Study Secondary Objective 3 Endpoints 5.3.1 Primary Endpoint 5.3.2 Secondary Endpoints 5.3.3 Exploratory Endpoints STUDY DESIGN AND DESCRIPTION | 17 |
| 5 | 3 Endpoints | 17 |
| | 5.3.1 Primary Endpoint | 17 |
| | 5.3.2 Secondary Endpoints. | 17 |
| | 5.3.3 Exploratory Endpoints | 17 |
| 6.0 | STODI DESIGNATION | |
| 6. | 1 Study Design | 19 |
| 6 | | |
| 6 | | |
| | 6.3.1 Rationale of Study Design | |
| | 6.3.2 Rationale for Dose | |
| | 6.3.3 Rationale for Endpoints | |
| | 6.3.4 Critical Procedures Based on Study Objectives: Timing of Procedures | 20 |
| 6.4 | | 20 |
| | Parameters | |
| 18 | , | 21 |
| 1, | <ul><li>6.5.1 Definition of Beginning of the Study.</li><li>6.5.2 Definition of End of the Study.</li></ul> | |
| | <ul><li>6.5.3 Definition of Study Completion</li><li>6.5.4 Definition of Study Discontinuation</li></ul> | |
| | • | |
| | <ul><li>6.5.5 Criteria for Premature Termination or Suspension of the Study</li><li>6.5.6 Criteria for Premature Termination or Suspension of a Site</li></ul> | |
| | 0.5.0 Chiena for Fremature reminiation of Suspension of a Site | 41 |

| 7.0 | SEL | ECTION AND DISCONTINUATION/WITHDRAWAL OF SUBJECTS | 22 |
|-----|-------|---------------------------------------------------------|-----|
| | 7.1 I | Excluded Medications, Supplements, Dietary Products | 22 |
| | 7.2 I | Diet, Fluid, Activity | 23 |
| | 7.2.1 | Diet and Fluid | 23 |
| | 7.2.2 | 2 Activity | Ø23 |
| | 7.3 | Criteria for Discontinuation or Withdrawal of a Subject | 23 |
| | 7.4 I | Criteria for Discontinuation or Withdrawal of a Subject | 24 |
| | 7.5 | Subject Replacement | 24 |
| 8.0 | CLI | NICAL STUDY MATERIAL MANAGEMENT | 25 |
| | 8.1 | Clinical Study Drug | 25 |
| | 8.1.1 | TAK-906 Capsule | 25 |
| | 8.1.2 | 2 Esomeprazole Capsule | 25 |
| | 8.1.3 | B Clinical Study Drug Labeling | 25 |
| | 8.1.4 | 4 Clinical Study Drug Inventory and Storage | 25 |
| | 8.1.5 | Clinical Study Drug Blinding | 25 |
| | 8.1.6 | 6 Randomization Code Creation and Storage | 26 |
| | 8.1.7 | 7 Clinical Trial Blind Maintenance/Unblinding Procedure | 26 |
| | 8.1.8 | | |
| 9.0 | | DY PROCEDURES | |
| | 9.1 | Administrative Procedures | 27 |
| | 9.1.1 | | |
| | 9.1.2 | | |
| | 9.1.3 | | |
| | 9.1.4 | 4 Concomitant Medications | 29 |
| | 9.2 | Clinical Procedures and Assessments | 29 |
| | 9.2.1 | 7.0 | |
| | 9.2.2 | 2 Height and Weight | 30 |
| | 923 | | 30 |
| | 9.2.4 | <b>C</b> | |
| 7, | 9.2.5 | | |
| 5) | 9.2.6 | | |
| | 9.2.7 | 2 | |
| | 9.2.8 | | |
| | 9.2.9 | 9 Clinical Laboratory Tests | 31 |
| | 9.3 I | PK Samples | 32 |

| 9.3.1 PK Measurements | 33 |
|---|---|
| 9.3.2 PK Measurements | 33 |
| 9.3.3 CCI | 34 |
| 9.3.4 Confinement | |
| 10.0 ADVERSE EVENTS | 35 |
| 10.1 Definitions and Elements of AEs 10.1.1 SAEs 10.1.2 Special Interest AEs | 35 |
| 10.1.1 SAEs | 37 |
| 10.1.2 Special Interest AEs | 38 |
| 10.2 AE Procedures 10.2.1 Assigning Severity/Intensity of AEs 10.2.2 Assigning Causality of AEs 10.2.3 Start Date 10.2.4 End Date 10.2.5 Pattern of Adverse Event (Frequency) 10.2.6 Action Taken With Study Treatment | 38 |
| 10.2.1 Assigning Severity/Intensity of AEs | 38 |
| 10.2.2 Assigning Causality of AEs. | 39 |
| 10.2.3 Start Date | 39 |
| 10.2.4 End Date | 40 |
| 10.2.5 Pattern of Adverse Event (Frequency) | 40 |
| 10.2.6 Action Taken With Study Treatment | 40 |
| 10.2.6 Action Taken With Study Treatment | 40 |
| 10.2.8 Collection and Reporting of AEs, SAEs, Special Interest AEs, and Abnormal | |
| LFTs | 41 |
| 11.0 STATISTICAL METHODS: | |
| 11.1 Statistical and Analytical Plans | |
| 11.1 Statistical and Analytical Flans 11.1.1 Analysis Sets | |
| 11.1.2 Analysis of Demography and Other Baseline Characteristics | |
| 11.1.3 PK Analysis | |
| 11.1.4 PD Analysis | |
| 11.1.5 Safety Analysis | |
| 11.2 Interim Analysis and Criteria for Early Termination | |
| 11.3 Determination of Sample Size | |
| 12.0 QUALITY CONTROL AND QUALITY ASSURANCE | |
| 2.1 Study-Site Monitoring Visits | |
| 12.2 Protocol Deviations | |
| 12.3 Quality Assurance Audits and Regulatory Agency Inspections | |
| 13.0 ETHICAL ASPECTS OF THE STUDY | |
| 13.1 IRB and/or IEC Approval | |
| 13.2 Subject Information, Informed Consent, and Subject Authorization | |
| 13.3 Subject Confidentiality | |

| Protocol Final | | 04 Feb 2019 |
|---|---|---|
| 13.4 Pu | ablication, Disclosure, and Clinical Trial Registration Policy | 50 |
| | Publication and Disclosure | |
| 13.4.2 | Clinical Trial Registration | 51 |
| 13.4.3 | Clinical Trial Results Disclosure | |
| 13.5 In: | INISTRATIVE AND REFERENCE INFORMATION dministrative Information Study Contact Information | 51 |
| 14.0 ADM | INISTRATIVE AND REFERENCE INFORMATION | |
| 14.1 Ac | dministrative Information | 52 |
| 14.1.1 | Study Contact Information | 52 |
| 14.1.2 | Investigator Agreement | 53 |
| 14.1.3 | Study-Related Responsibilities | 54 |
| 14.1.4 | List of Abbreviations | 55 |
| 15.0 DATA | A HANDLING AND RECORDKEEPING | 57 |
| 15.1 CI | RFs (Electronic and/or Paper) | 57 |
| 15.2 Re | ecord Retention | 57 |
| 16.0 REFE | RENCES | 59 |
| 17.0 APPE | NDICES | 60 |
| LIST OF IN- | Study Contact Information Investigator Agreement Study-Related Responsibilities List of Abbreviations A HANDLING AND RECORDKEEPING RFs (Electronic and/or Paper) ecord Retention RENCES NDICES Study Drugg Planned Dood ovels | |
| Table 6.a | Study Drugs Planned Dose Levels | 19 |
| Table 7.a | Excluded Medications, Supplements, and Dietary Products | 22 |
| Table 9.a | Primary Specimen Collections | |
| Table 10.a | Takeda Medically Significant AE List | 38 |
| | GOV. | |
| LIST OF IN- | TEXT FIGURES | |
| Figure 2.a | Schematic of Study Design | 10 |
| | Schematics of Single-Sequence Design | |
| >Q. | | |
| LIST OF AP | PENDICES | |
| Appendix A | Responsibilities of the Investigator | 61 |
| Appendix B | Elements of the Subject Informed Consent | 63 |
| Appendix C | Investigator Consent to the Use of Personal Information | 66 |
| Appendix D | Pregnancy and Contraception | 67 |

### 1.0 STUDY SUMMARY

| Millennium Pharmaceuticals, Inc. a wholly owned subsidiary of Takeda Pharmaceutical Company, Ltd 40 Landsdowne Street | Compound:<br>TAK-906 | 1 St |
|---|---|---|
| Cambridge, Massachusetts USA 02139 Study Identifier: TAK-906-1006 (CA27239) | Phase: 1 | |

**Protocol Title**: A Single-Sequence, Open-Label, 2-Period, Crossover Study to Evaluate the Effect of the Proton Pump Inhibitor Esomeprazole on the Single-Dose Pharmacokinetics of Oral TAK-906 in Healthy Adult Subjects

### **Study Design:**

This is a single-sequence, open-label, 2-period, crossover study in 12 healthy adult subjects. The study is designed to investigate the effect of a proton pump inhibitor (PPI) esomeprazole on the PK of TAK-906.

The study will include a Screening Visit, Study Period 1 (Days 1 to 3), followed by at least a 4-day washout (from the time of TAK-906 dose on Day 1), Study Period 2 (Days 1 to 6), and finally a Follow-up Visit.

In Study Period 1, subjects will be confined from the day prior to dosing (Day -1), at the time indicated by the Clinical Research Unit (CRU), until after the 48-hour blood draw (Day 3). In Study Period 2, subjects will come to the CRU on the mornings of Day 1 and Day 2, at the time indicated by the CRU, for dosing and/or study procedures as appropriate. Subjects will be confined from morning of Day 3, at the time indicated by the CRU, until after the 48-hour blood draw on Day 6. At any time, a subject may be required to remain at the CRU for longer at the discretion of the Investigator.

On Day 1 of Study Period 1, subjects will receive a single oral dose of TAK-906. On Days 1 through 5 of Study Period 2, subjects will receive esomeprazole dose once daily (QD). On Day 4 of Study Period 2, a single oral dose of TAK-906 will be administered 1 hour following the esomeprazole dose. Serial blood samples will be collected predose and for 48 hours after each TAK-906 dose to determine the pharmacokinetics (PK) of TAK-906.

There will be a washout of at least 4 days between dosing in Study Period 1 and first dosing in Study Period 2.

All subjects who received at least one dose of study drug (including subjects who terminate the study early) will return to the Clinical Research Unit (CRU) approximately 10-14 days after the last dose of TAK-906 for follow-up procedures, and to determine if any adverse event (AE) has occurred since the last study visit.

- Study Primary Objective:
- To evaluate the effect of the PPI esomeprazole on the single-dose PK of orally (PO) administered TAK-906.
- Secondary Objectives:
- To evaluate the safety and tolerability of a single PO dose of TAK-906 in the presence and absence of the PPI esomeprazole.

**Study Subject Population:** Males and females (with no childbearing potential) aged 18 to 55 years, inclusive, at the Screening Visit. Body mass index (BMI)  $\geq$ 18.0 and  $\leq$ 30.0 kg/m<sup>2</sup> at screening.

| Planned Number of Subjects: | Planned Number of Sites: |
|---|---|
| 12 | 1 |
| Dose Levels: | Route of Administration: |
| Study Period 1 (Treatment A): | Oral |
| 25 mg TAK-906 (1 x 25 mg TAK-906 capsule) | |
| Study Period 2 (Treatment B): | |
| 40 mg esomeprazole (1 x 40 mg NEXIUM <sup>®</sup> capsule, or generic equivalent) | |
| 25 mg TAK-906 (1 x 25 mg TAK-906 capsule) | |

Riobe

### **Duration of Treatment:**

On Day 1 of Study Period 1, subjects will receive a single oral dose of TAK-906.

On Days 1 through 5 of Study Period 2, subjects will receive QD doses of esomeprazole. On Day 4 of Study Period 2, subjects will receive a single oral dose of TAK-906 1 hour following esomeprazole dose.

### **Planned Study Duration:**

le Leine Of I Approximately 50 days including Screening Period

### **Main Criteria for Inclusion:**

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study.

- 1. Healthy, adult, male or female, 18-55 years of age, inclusive, at screening.
- 2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study, based on screening urine cotinine test.
- 3. Body mass index (BMI)  $\geq 18.0$  and  $\leq 30.0$  kg/m<sup>2</sup> at screening.
- 4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiographs (ECGs), as deemed by the Investigator or designee.
- 5. For a male or female of non-childbearing potential, use acceptable birth control methods as indicated in Appendix D.
- 6. A male subject who is nonsterilized and sexually active with a female partner of childbearing potential must agree to use a barrier method of contraception from the signing of informed consent form (ICF) throughout the duration of the study and through to the follow up (ie, 10-14 days after the last dose of TAK-906) (refer to Appendix D).
- 7. If male, must agree not to donate sperm from the first dosing until follow-up visit (ie, 10-14 days after the last dose of TAK-906) (refer to Appendix D).
- 8. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

### **Main Criteria for Exclusion:**

The subject must be excluded from participating in the study if the subject:

- 1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
- 2. History or presence of clinically significant endocrine, gastrointestinal (including motility disorder and intestinal obstruction), cardiovascular, hematological, hepatic, immunological, renal, respiration, genitourinary, or major neurological (including stroke and chronic seizures) or any other clinically significant abnormalities or disease in the opinion of the Investigator or designee.
- 3. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
- 4. History of cancer (malignancy).
- 5. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
- 6. History or presence of hypersensitivity or idiosyncratic reaction to TAK-906 or related compounds, or to esomeprazole or PPIs (see NEXIUM® US product insert [USPI]).
- Female subjects of childbearing potential.
- Female subjects with a positive pregnancy test or who is lactating.
- Positive urine drug or alcohol results at screening or first check-in.
- 10. Positive urine cotinine at screening.
- 11. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).

- 12. QTcF interval is >450 msec or ECG findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
- 13. Estimated creatinine clearance <90 mL/min at screening.
- 14. Unable to refrain from or anticipates the use of:
  - Any drug, including prescription and non-prescription medications (including PPIs, antacids, and H<sub>2</sub>-antagonist), herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Thyroid hormone replacement medication may be permitted if the subject has been on the same stable dose for the immediate 3 months prior to first study drug administration. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the Investigator or designee.
  - Any drugs known to significantly affect the absorption, distribution, metabolism, or elimination of study drugs (TAK-906 or esomeprazole) within 28 days prior to the first dosing and throughout the study. Appropriate sources (eg, Flockhart Table<sup>TM</sup>) will be consulted to confirm lack of PK/pharmacodynamic interaction with study drug.
- 15. Has been on a diet incompatible with the on-study diet, in the opinion of the **Investigator** or designee, within the 30 days prior to the first dosing and throughout the study.
- 16. Donation of blood or significant blood loss (eg, approximately 500 mL) within 56 days prior to the first dosing.
- 17. Plasma donation within 7 days prior to the first dosing.
- 18. Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Study Period 1 of the current study.

### Main Criteria for Evaluation and Analyses:

The primary endpoint of the study is:

The following plasma PK parameters for TAK-906 on Day 1 in Study Period 1 and on Day 4 in Study Period 2:

- C<sub>max</sub>: Maximum observed concentration.
- AUC<sub>last</sub>: Area under the concentration-time curve from time 0 to time of the last quantifiable concentration.
- AUC<sub>inf</sub>: Area under the concentration-time curve from time 0 to infinity.

The secondary endpoints include the following:

- Treatment emergent adverse event (TEAE) assessments.
- Vital signs.
- 12-lead ECG.
- Clinical laboratory testing (hematology, serum chemistry and urine analysis).

CC

150 USE

### **Statistical Considerations:**

For evaluation of potential effect of esomeprazole on TAK-906 PK, an ANOVA will be performed on the In-transformed C<sub>max</sub>, AUC<sub>last</sub>, and AUC<sub>inf</sub>. The ANOVA model will include treatment as fixed effect and subject as a random effect. Each ANOVA will include calculation of least-squares means (LSM) as well as the difference between treatment LSM. The geometric mean of the relative bioavailability of the TAK-906 with esomeprazole regimen relative to the TAK-906 regimen alone and the associated 90% CIs will be determined by exponentiation of the appropriate estimates for the difference between regimens in the log-transformed parameters.

### **Sample Size Justification:**

A total of twelve (12) subjects will be enrolled in this study. This sample size will provide at least 80% power to conclude the C<sub>max</sub> of TAK-906 will not decrease more than 50% in the presence of esomeprazole, assuming that the intra-subject %CV for C<sub>max</sub> of TAK-906 will not exceed 45% and a true ratio of 0.8. Lower intra-subject variability was observed for AUC in previous studies; therefore, the power is expected to be greater for AUC.

A. Lo oe greate, on wand subject to property of Takeda. For noncommercial use only and subject to property of Takeda.

### 2.0 STUDY SCHEMATIC

### Figure 2.a Schematic of Study Design

| Screening | Study Period 1 <sup>a</sup> | | |
|---|---|---|---|
| | Day -1 | Day 1 | Days 2 - 3 |
| Within Day -28 to -2 for screening; first | Check-in | TAK-906 Dosing | 2010 |
| dosing in Study Period 1 | | Plasma sampling for TAK-906 PK and safety monitoring for at least 48 hours postdose | |
| | < Confinement b, c | | |

<sup>&</sup>lt;sup>a</sup> There will be a washout of at least 4 days between dosing in Study Period 1 and first dosing in Study Period 2.

<sup>b</sup> A subject may be required to remain at the CRU for longer at the discretion of the Investigator or designee.

<sup>&</sup>lt;sup>c</sup> Subjects will start the confinement on Day -1 of Study Period 1 and be released from CRU after Day 3 study assessments are complete. In Study Period 2, subjects will return to the CRU on the morning of Days 1 and 2 for dosing and/or study procedures as appropriate. Subjects will be confined from morning of Day 3 of Study Period 2, at the time indicated by the CRU, until after 48-hour blood draw on Day 6.

| | Treatn | nent Study Period 2 a | 20 | | Study exit | Follow-up b |
|---|---|---|---|---|---|---|
| Days 1-2 | Day 3 | Day 4 | | | | |
| | Check-in | Oll | Day 6 of | 10.14 days | | |
| Esomeprazole dosing | Esomeprazole dosing | Esomeprazole dosing TAK-906 Dosing | Esomeprazole dosing | | Treatment<br>Study | 10-14 days<br>after last<br>dosing |
| | | Plasma sampling for TA monitoring for at least 4 | Period 2 | ucomg | | |
| Outpatient visit | < | | | | | |

<sup>&</sup>lt;sup>a</sup> There will be a washout of at least 4 days between dosing in Study Period 1 and first dosing in Study Period 2. <sup>b</sup> All subjects who received at least one dose of study drug (including subjects who terminate the study early) will return to the CRU approximately 10-14 days after the last dose of TAK-906 for follow-up procedures, and to determine if any AE has occurred since the last study visit

as appropriate. Subjects will be confined from morning of Day 3 of Study Period 2, at the time indicated by the CRU, until after 48-hour blood draw on Day 6.

<sup>&</sup>lt;sup>c</sup> A subject may be required to remain at the CRU for longer at the discretion of the Investigator or designee.

<sup>d</sup> In Study Period 2, subjects will return to the CRU on the morning of Days 1 and 2 for dosing and/or study procedures

**Schematics of Single-Sequence Design** Figure 2.b



## 3.0 SCHEDULE OF STUDY PROCEDURES

| | Screening | | Study 1 | Period 1 | (a) | | | | Study P | eriod 2 | $\mathcal{V}$ | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day -28 to -2 | | Day | | Day | | | | | | 10-14 days after last dose of TAK-906 | | |
| | - | | Predose | | | | | | 3/0 | 0 | | | |
| Procedures/Assessments | | -1 | (Day 1) | 1 | 2 | 3 | 1 | 2 | 3 | 4 | 5 | 6 | |
| Administrative Procedures | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | * | 0 | | | | | |
| Medical history/demographics | X | | | | | | ./0 | | | | | | |
| Prior and concomitant medication | | | | | | Co | ntinuous l | Monite | oring | | | | |
| review | | | | | | | iitiiiuous i | vioiiiu | Jing | | | | |
| Clinical Procedures/Assessments | | | | | | _ ^ | <i>)</i> | | | | | | |
| Full physical examination | X | | X (b) | | | 0 | | | | | | | X |
| Height | X | | | | 1 | ) | | | | | | | |
| Weight | X | | | | | | | | | | | | |
| BMI | X | | | | Ó | | | | | | | | |
| 12-Lead Safety ECG | X | | X (c), (b) | $X^{(c)}$ | ) | X | | | | X (c) | | X (h) | X |
| Supine vital signs (heart rate, systolic | X | | X (c),(b) | X (c) | | X | | | | X (c) | | X (h) | X |
| blood pressure and diastolic blood | | | | | | | | | | | | | |
| pressure) | | | | ) | | | | | | | | | |
| Vital signs (respiratory rate, oral [at the | X | | X(O) | | | | | | | | | | |
| floor of the mouth]/tympanic | | | ~0°. | | | | | | | | | | |
| temperature) | | | <i>d</i> , | | | | | | | | | | |
| TAK-906 administration <sup>(d)</sup> | | _< | | X | | | | | | X | | | |
| Esomeprazole administration (e) | | <u>Q</u> | | | | | X | X | X | . X | X | | |
| AE monitoring | | <u></u> | | | | | Cont | inuous | s Monito | oring | | | |
| <b>Laboratory Procedures/Assessments</b> | | | | • | | • | 4.5 | | • | | , | - 45 | |
| Hematology | X | X | | | | | X (b) | | | | | X (h) | X |
| Urinalysis | X | X | | | | | X (b) | | | | | X (h) | X |
| Chemistry | √X | X | | | | | X (b) | | | | | X (h) | X |
| Serum Pregnancy Test (♀only) | X | X | | | | | | | | | | | |
| Serum FSH (PMP $\stackrel{\frown}{}$ only) | X | | | | | | | | | | | | |
| Urine drug screen | X | X | | | | | X | | | | | | |
| Urine alcohol test (f) | X | X | | | | | X | | | | | | |
| Urine cotinine test | X | | | | | | | | | | | | |

| | | | ~ | | (a) | | 1 | | | | - | $\sim$ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | Study I | Period 1 | (a) | | Study Period 2 | | | | | | Follow-up |
| | | | | | | | | | | | | | 10-14 days after last dose of |
| | Day -28 to -2 | | 1 | Day | | | | | Da | ıy 🧷 | 16. | | TAK-906 |
| | | | Predose | | | | | | | 0 | <b>*</b> | | |
| Procedures/Assessments | | -1 | (Day 1) | 1 | 2 | 3 | 1 | 2 | 3 | 0,4 | 5 | 6 | |
| Hepatitis screen | X | | | | | | | | 1/4 | | | | |
| Human immunodeficiency virus (HIV) | X | | | | | | | , | .0 | | | | |
| Pharmacokinetics Evaluations | | | | | | | | × | 0 | | | | |
| Blood for plasma TAK-906 (g) | | | X | | ] | X | XX | | | | X | | |
| CCI | | | | | | | | O | | | | | |
| CCI | | | | | | | | | | | | | |
| Other | | | | | | | | | | | | | |
| Confinement | | | X | X | - | 5 | | | | X | X | | |
| Returns (i) | | | | | | | X | X | | | | | |
| Meals fasting | | | X | X | | (Q) | X | X | X | X | X | | |

- (a) There will be a minimum 4-day washout between Study Periods 1 and 2, starting from administration of TAK-906 on Day 1 of Study Period 1.
- (b) Day 1 predose assessment may be done within approximately 24 hours prior to study drug administration.
- (c) Measured predose and at 1, 2, 4, 8, and 48 hours postdose (times relative to TAK-906 dose). Subjects should have rested in a supine position for at least 5 minutes before the measurements.
- (d) Both doses of TAK-906 (Day 1 of Study Period 1 and Day 4 of Study Period 2) will be administered after an overnight fast of at least 10 hours and subjects will be required to fast for at least 4 hours postdose. For Study Period 2, TAK-906 will be administered I h after esomeprazole dose on Day 4.
- (e) Esomeprazole will be administered once daily at the same time each day and 1 hour prior to TAK-906 on Day 4. On Days 1 to 3 and Day 5, subjects will be required to fast for at least 1 hour prior to esomeprazole dosing and to remain fasting for at least 2 hours postdose.
- (f) An alcohol breath test may be performed at the discretion of the Investigator.
- (g) Blood samples for TAK-906 assay will be collected on Day 1 of Study Period 1 and Day 4 of Study Period 2 predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose (times relative to TAK-906 dose). The 16-hour postdose on Day 1 of Study Period 1 and Day 4 of Study Period 2 will be either on Day 1 or Day 2 of Period 1 and Day 4 or Day 5 of Study Period 2, depending on the time of dosing on Day 1 of Study Period 1 and Day 4 of Study Period 2, respectively.
- (h) To be performed on Day 6 of Study Period 2 or prior to early termination from the study.
- (i) Subjects will return to the CRU every morning on Days 1 and 2 of Study Period 2 to receive the esomeprazole dosing (± 1 hour of Day 1 dosing).

Abbreviations:  $\bigcirc$  = Female, AE = Adverse events, **BMI** = Body mass index, CRU = Clinical research unit, DNA = Deoxyribose nucleic acid, ECG = Electrocardiogram, HIV = Human immunodeficiency virus, PMP = **Postmenopausal**, PK = Pharmacokinetics.

Background for TAK-906

The intended indication for TAK-906 is to treat patients with gastroparesis, a disorder of the stomach characterized by delayed gastric emptying in the absence of mechanical obstruction Symptoms are chronic with episodic symptom exacerbation [1]. These symptoms are chronic with episodic symptom exacerbation [1]. These symptoms are chronic with episodic symptom exacerbation [1]. These symptoms are chronic with episodic symptom exacerbation [1]. These symptoms are chronic with episodic symptom exacerbation [1]. These symptoms are chronic with episodic symptom exacerbation [1]. cases of chronic gastroparesis, diabetic (29%), postsurgical (13%), and idiopathic (36%) etiologies comprise the majority of cases in the tertiary referral setting [3].

TAK-906 is a peripherally selective (ie, very limited penetration of the blood brain barrier [BBB]) dopamine D2/D3 receptor antagonist. It demonstrated suitable PK and PD activity in a phase 1 study and other completed studies. Therefore TAK-906 is expected to reduce nausea and vomiting, without the side effects which restrict the use. Because of its low BBB penetration and a weak human ether-a-go-go-related gene (hERG) channel affinity indicative of a low potential cardiac risk, TAK-906 is anticipated to have an improved safety **profile**, compared to other D2/D3 antagonist (eg., metoclopramide and domperidone).

The solubility of TAK-906 is pH dependent (decreases with the increase of pH), and it is classified as a Biopharmaceutical Classification System class IV drug. Studies of in vitro metabolism suggest that TAK-906 is mainly metabolized by CYP2C8 and CYP3A4/5,

The relative contribution ratio of CYP and non-CYP toward in vitro metabolism of TAK-906 using human hepatic S9 cell line was 43.3% and 56.7%, respectively. TAK-906 is also a substrate of P-glycoprotein (P-gp), organic anion-transporting polypeptide (OATP)1B1 and OATP1B3.

TAK-906 shows rapid absorption and rapid elimination. Median  $T_{max}$  was 1.1 hours postdose. The half-life (T½) following a single PO dose averaged approximately 4 hours when administered in the fasted state. Following administration of single PO doses of TAK-906 maleate between 5 and 300 mg, exposure to TAK-906 increased in a manner generally proportional to dose increment. Food had a significant impact on reducing the exposure to TAK-906 in healthy subjects. Coadministration of itraconazole 200 mg for 5 days with TAK-906 maleate increased TAK-906 mean C<sub>max</sub> by approximately 2.0-fold and AUCinf by approximately 1.3-fold. TAK-906 is not classified as a sensitive CYP3A4 substrate.

Refer to the Investigator's Brochure (IB) for detailed background information on TAK-906 [4].

### **Background for Esomeprazole**

Esomeprazole, the S-enantiomer of omeprazole, is a PPI that inhibits gastric acid secretion by suppressing H+ ion formation through inhibition of the H+/K+ ATPase enzyme system at the secretory surface of gastric parietal cells. Esomeprazole is indicated for the treatment of heartburn and other symptoms associated with gastroesophageal reflux disease and, in combination with

clarithromycin and amoxicillin, for the eradication of Helicobacter pylori. The recommended adult dosages are 20 mg to 40 mg QD, administered at least one hour before meals [5].

After oral administration of esomeprazole capsule formulation,  $C_{max}$  occurs at approximately 1.5 hours ( $T_{max}$ ). At repeated QD dosing with 40 mg, the systemic bioavailability is approximately 90% compared to 64% after a single dose of 40 mg [5]. The administration of food with esomeprazole reduces AUC and  $C_{max}$  by 43 to 53% and 33 to 53%, respectively; however this does not have a significant influence on the effect of esomeprazole on intra-gastric acidity [6]. Esomeprazole is 97% bound to plasma proteins [5]. Esomeprazole is acid-labile and rapidly degrades under acidic conditions, but is very stable in alkaline media. Esomeprazole has been shown to be optically stable and the degree of inversion to be negligible [5].

Esomeprazole is extensively metabolized in the liver (to a lesser extent than racemic omeprazole), primarily by CYP2C19 and CYP3A to form the hydroxy, desmethyl, and sulfone metabolites. None of the identified metabolites exhibit any of the significant anti-secretory effects displayed by the parent drug [5].

Elimination of the drug is rapid with a terminal elimination half-life of about 1.3 hours. Approximately 80% of an oral dose of esomeprazole is excreted as inactive metabolites in the urine, and 20% in feces. Less than 1% of the parent drug is excreted unchanged in the urine [5].

The most common adverse reactions associated with esomeprazole administration are: headache, abdominal pain, constipation, diarrhea, flatulence, nausea, and dry mouth [5].

## 4.3 Rationale for the Proposed Study

The solubility of TAK-906 is pH dependent (decreases with the increase of pH). PPIs are commonly used by gastroparesis patients to relieve symptoms of gastroesophageal reflux such as heartburn or regurgitation that frequently overlap with gastroparesis. This group of agents suppresses gastric acid secretion by specific inhibition of the H<sup>+</sup>/K<sup>+</sup>-ATPase pump in gastric parietal cells, thereby increasing gastric pH for a sustained time, and thus may alter the bioavailability of drugs with pH-dependent solubility when used together.

Esomeprazole is widely prescribed. It is known to have a strong anti-secretory effect, suppressing the production of gastric acid from parietal cells, and increasing pH. Esomeprazole is expected to lack the potential to interact directly with TAK-906, for example through CYP3A4 metabolic interaction [7]. In addition, esomeprazole has a good safety and tolerability profile, and was found to be well-tolerated in healthy volunteers [8].

### 4.4 Benefit/Risk Profile

The dose of TAK-906 administered in this study is not anticipated to induce any potential risk or benefit to subjects participating in this study. Based on the first-in-human phase 1 study, a single dose of 25 mg TAK-906 is expected to be well tolerated.

The dose of esomeprazole administered in this study is not anticipated to induce any potential risk or benefit to subjects participating in this study, and it is administered according to the dosing recommendations found in the full prescribing information for NEXIUM<sup>®</sup> [5].

.a employed by this protocol (ie, 12-lead ECG, vital signing, and physical examination) are adequate to protect the all TEALS.

.t health benefit for study participants from receipt of study drug. An are healthly subjects enrolled in this study is the free medical tests received, arring the study.

arring the study.

An are healthly subjects enrolled in this study is the free medical tests received, arring the study.

An are healthly subjects enrolled in this study is the free medical tests received, arring the study.

An are healthly subjects enrolled in this study is the free medical tests received, arring the study.

An are healthly subjects enrolled in this study is the free medical tests received, arring the study. There will be no direct health benefit for study participants from receipt of study drug. An indirect health benefit to the healthy subjects enrolled in this study is the free medical tests received at screening and during the study.

### 5.0 STUDY OBJECTIVES AND ENDPOINTS

### 5.1 Hypothesis

NA

## 5.2 Study Objectives

## 5.2.1 Study Primary Objective

• To evaluate the effect of the PPI, esomeprazole, on the single-dose PK of PO administrated TAK-906.

## 5.2.2 Study Secondary Objective

• To evaluate the safety and tolerability of a single PO dose of TAK-906 in the presence and absence of the PPI, esomeprazole.

### 5.3 Endpoints

### 5.3.1 Primary Endpoint

The primary endpoint of the study is:

The following plasma PK parameters for TAK-906 on Day 1 in Study Period 1 and on Day 4 in Study Period 2

- C<sub>max</sub>: Maximum observed concentration.
- AUC<sub>last</sub>: Area under the concentration-time curve from time 0 to time of the last quantifiable concentration.
- AUC<sub>inf</sub>: Area under the concentration-time curve from time 0 to infinity.

## 5.3.2 Secondary Endpoints

Secondary endpoints include:

- TEAE assessments.
- Vital signs.
- 12-lead ECG.
- Clinical laboratory testing (hematology, serum chemistry, and urine analysis).

### 5.3.3 Exploratory Endpoints

CCI



Properly of Takeda. For non-commercial use only and subject to the applica

This is a single-sequence, open-label, 2-period crossover study in 12 healthy adult subjects. The study is designed to investigate the effect of a PPI esomeprazole on the PK of TAK-906

The study will include a Screening Visit, a Study Period 1 (F)

4-day washout from the time of Take-906 Visit.

Screening of subjects will occur within 28 days prior to the first dosing.

In Study Period 1, subjects will be confined from the day prior to dosing (Day -1), at the time indicated by the CRU, until after the 48-hour blood draw (Day 3). In Study Period 2, subjects will come to the CRU on the mornings of Day 1 to Day 2, at the time indicated by the CRU, for dosing and/or study procedures as appropriate. Subjects will be confined from morning of Day 3, at the time indicated by the CRU, until after the 48-hour blood draw on Day 6. At any time, a subject may be required to remain at the CRU for longer at the discretion of the Investigator.

On Day 1 of Study Period 1, subjects will receive a single oral dose of TAK-906. On Days 1 through 5 of Study Period 2, subjects will receive esomeprazole dose QD. On Day 4 of Study Period 2, a single oral dose of TAK-906 will be administered 1 hour following the esomeprazole dose. Serial blood samples will be collected predose and for 48 hours after each TAK-906 dose to determine the PK of TAK-906.

There will be a washout of at least 4 days between dosing in Study Period 1 and first dosing in Study Period 2.

All subjects who received at least one dose of study drug (including subjects who terminate the study early) will return to the CRU approximately 10-14 days after the last dose of TAK-906 for follow-up procedures, and to determine if any AE has occurred since the last study visit.

Please refer to Section 2.0 for study schematics.

The planned dose levels of TAK-906 and esomeprazole to be used are outlined in Table 6.a.

Study Drugs Planned Dose Levels Table 6.a

| 1890. | Dose | Route of Administration |
|------------------------------|-------|-------------------------|
| Study Period 1 (Treatment A) | | |
| TAK-906 | 25 mg | Oral capsule |
| Study Period 2 (Treatment B) | | |
| TAK-906 | 25 mg | Oral capsule |
| Esomeprazole | 40 mg | Oral capsule |

### 6.2 **Dose Escalation**

NA

## 6.3 Rationale for Study Design, Dose, and Endpoints

### 6.3.1 Rationale of Study Design

This is a single-sequence, open-label, 2-period crossover study.

An open-label design was employed in this study, since the primary objective is to assess PK and it is unnecessary to be blinded.

Since esomeprazole may have a prolonged effect on acid secretion due to its irreversible binding to H+/K+ ATPase pump, a single-sequence design in which esomeprazole is administered in Study Period 2 was selected to ensure that there is no carryover pharmacodynamic effect on gastric acid secretion for the reference treatment (TAK-906 alone).

The washout period between TAK-906 doses in each period is considered sufficient to ensure minimal carryover effects of the TAK-906.

### **6.3.2** Rationale for Dose

**TAK-906:** Based on the first-in-human phase 1 study, administration of single PO doses of TAK-906 maleate ranging from 5 to 300 mg have been well-tolerated in healthy men and women. Overall, the incidence of TEAEs was low in the study. There were no SAEs or severe AEs reported during the study, and no subjects discontinued due to an AE. Based on the results of the clinical studies, 25 mg dose of TAK-906 is expected to be the clinically efficacious dose that is well below the maximum tested dose of 300 mg.

**Esomeprazole:** A dose of 40 mg esomeprazole daily is within the recommended dose as prescribed in the labeling [5]. In addition, multiple doses will ensure maximum inhibition of acid secretion by esomeprazole [6]. The maximum recommended dose of esomeprazole (40 mg per day) was selected to ensure that any possible PK interactions are detected.

## **6.3.3** Rationale for Endpoints

The primary PK endpoints will include  $C_{max}$ ,  $AUC_{inf}$  and  $AUC_{last}$ , as these parameters describe the exposure and bioavailability of TAK-906 and are the most relevant PK parameters for the purpose of evaluating an interaction.

## 6.3.4 Critical Procedures Based on Study Objectives: Timing of Procedures

For this study, the blood collection for plasma concentrations for TAK-906 is the critical procedure and samples are required to be collected, as appropriate, as close to the scheduled times defined in this protocol as possible.

# 6.4 Study Design/Dosing/Procedures Modifications Permitted Within Protocol Parameters

The dose and administration of the study drugs to any subject may not be modified. If necessary a subject must be discontinued for the reasons described in Section 6.5.5.

The beginning of the study will be defined as the beginning of the screening (ie, signing of the ICF) of the first subject.

6.5.2 Definition of End of the Study

The end of

The end of study is defined as the date of the last scheduled study procedure as outlined in the Schedule of Study Procedures (Section 3.0).

### **6.5.3** Definition of Study Completion

The end of the study is defined as the completion of the evaluations in the follow-up visit for the last subject in the study.

This time period may change in the event that the study is terminated early or the last subject is lost to follow-up.

### 6.5.4 Definition of Study Discontinuation

In consultation with the Sponsor, Celerion reserves the right to terminate the study in the interest of subject welfare.

The Sponsor reserves the right to suspend or terminate the study at any time.

### 6.5.5 Criteria for Premature Termination or Suspension of the Study

The study will be completed as planned unless one or more of the following criteria are satisfied that require temporary suspension or early termination of the study:

- New information or other evaluation regarding the safety or efficacy of the study medication that indicates a change in the known risk/benefit profile for the product, such that the risk is no longer acceptable for subjects participating in the study.
- Significant violation of Good Clinical Practice (GCP) that compromises the ability to achieve the primary study objectives or compromises subject safety.

### Criteria for Premature Termination or Suspension of a Site

Excluded Medications, Supplements, Dietary Products

Concomitant medications will be prohibited as listed in the exclusion criteria in Section 9.1.2.22

After the first dose, acetaminophen (up to 2 g per 24 hour period) may be administered at the discretion of the Investigator or designee. Thyroid hormone replacement is study drug administration

If deviations occur, the investigator or designee in consultation with the Sponsor if needed will decide on a case-by-case basis whether the subject may continue participation in the study.

All medications taken by subjects during the course of the study will be recorded.

Use of excluded agents (prescription or non-prescription) or dietary products is outlined in Table 7.a.

**Excluded Medications, Supplements, and Dietary Products** Table 7.a

| Category | Between Screening and First Dosing (Days -28 to predose [Day 1]) | Post First Dosing (Day 1) to Follow-Up |
|---|---|---|
| Alcohol | Prohibited from 48 hours prior to first dosing | Prohibited from 48 hours prior to first dosing in each period and throughout until end of PK collection in Treatment Period 2. |
| Xanthine and/or caffeine | Prohibited from 24 hours prior to first dosing a | Prohibited from 24 hours prior to first dosing in each period and throughout the period of PK sample collection in each Study Period a. |
| Nicotine | Prohibited from 3 months prior to first dosing | Prohibited from 3 months prior to first dosing in each period until end of PK collection in Study Period 2 |
| Medications | See Sections 7.1 and 9.1.2.2 | See Sections 7.1 and 9.1.2.2 |
| Food substance | | |
| Grapefruit/Seville orange | Prohibited from 14 days prior to first dosing | Prohibited until end of PK collection in Treatment Period 2. |
| Other Fruit Juice | Prohibited from 72 hours prior to first dosing | Prohibited from 72 hours prior to first dosing in each period and throughout the period of PK sample collection in each Study Period. |
| Vegetables from the mustard green<br>family (eg, kale, broccoli,<br>watercress, collard greens, kohlrabi,<br>Brussels sprouts, mustard), and<br>charbroiled meats | Prohibited from 7 days prior to first dosing | Prohibited until end of PK collection in Study Period 2. |

small amounts of caffeine derived from normal foodstuffs eg, 250 mL/8 oz./1 cup decaffeinated coffee or other decaffeinated beverage, per day, with the exception of espresso; 45 g/1.5 oz. chocolate bar, per day, would not be considered a deviation to this restriction.

Water (except water provided with each oral dosing) will be restricted 1 hour prior to and 1 hour after each oral study drug administration, but will be allowed ad libitum at all other times when dosing occurs at the CRU. Other fluids may be given as part of most restricted at all other times throughout the

On Day 1 of Study Period 1 and Day 4 of Study Period 2, subjects will fast overnight for at least 10 hours prior to TAK-906 administration and will continue to fast for at least 4 hours postdose.

On Days 1 to 3 and Day 5 of Study Period 2, subjects will fast for at least 1 hour prior to dosing and will continue to fast for at least 2 hours postdose.

When confined, standard meals and snacks will be provided at appropriate times, except when they are required to fast. When confined in the CRU, subjects will be required to fast from all food and drink except water between meals and snacks.

Each meal and/or snacks served at the CRU will be standardized and will be similar in caloric content and composition and will be taken at approximately the same time in each treatment period.

## 7.2.2 Activity

Subjects will remain ambulatory or seated upright for the first 4 hours postdose, except when they are supine or semi-reclined for study procedures. However, should AEs occur at any time, subjects may be placed in an appropriate position or will be permitted to lie down on their right side.

Subjects will be instructed to refrain from strenuous physical activity which could cause muscle aches or injury, including contact sports at any time from screening until completion of the study.

### 7.3 Criteria for Discontinuation or Withdrawal of a Subject

Subjects are free to withdraw from the study at any time for any reason.

In addition, subjects may be withdrawn from the study by the Investigator or designee for the following reasons:

- Difficulties in blood collection.
- Positive pregnancy test.
- Positive drug and alcohol test.

A subject may be withdrawn by the Investigator (or designee) or the Sponsor if enrollment into the study is inappropriate, the study plan is violated, or for administrative and/or other safety reasons.

### Procedures for Discontinuation or Withdrawal of a Subject 7.4

The investigator may discontinue a subject's study participation at any time during the study when the subject meets the study termination criteria described in Section 7.3. In addition, a subject may discontinue his or her participation without giving a reason at any time during the study. Should a subject's participation be discontinued, the primary criterion for termination must be recorded by the Investigator. In addition, efforts should be made to perform all procedures scheduled for the follow-up or early termination as described in Section 3.0.

### 7.5 **Subject Replacement**

 and subject to Subjects who discontinue for non-safety reasons may be replaced at the discretion of the Investigator in consultation with the Sponsor. Subjects who discontinue for safety reasons will not

### 8.0 CLINICAL STUDY MATERIAL MANAGEMENT

### 8.1 Clinical Study Drug

### **8.1.1** TAK-906 Capsule

A single 25 mg dose of TAK-906 maleate capsule will be administered on Day 1 of Study Period 1 and on Day 4 of Study Period 2 of the study.

Oral dose of TAK-906 drug product is a nonsterile, capsule dosage form, supplied in a hard gelatin capsule of TAK-906 maleate. TAK-906 maleate is the active pharmaceutical ingredient. No other active ingredients are included in the drug product.

### 8.1.2 Esomeprazole Capsule

Once-daily (QD) 40 mg dose of esomeprazole capsules (Nexium® capsule, or generic equivalent) will be administered on Days 1 through 5 of Study Period 2.

Oral dose of esomeprazole drug product is a nonsterile, capsule dosage form, supplied in a hard gelatin capsule of esomeprazole. Esomeprazole is the active pharmaceutical ingredient. No other active ingredients are included in the drug product.

## 8.1.3 Clinical Study Drug Labeling

TAK-906 capsule containers will be affixed with a clinical label in accordance with local regulatory requirements.

Esomeprazole capsule will be provided with the commercially available package and labeling in accordance with local regulatory requirements.

### 8.1.4 Clinical Study Drug Inventory and Storage

The Sponsor will supply sufficient quantities of TAK-906 products to allow completion of this study.

Celerion will provide sufficient quantities of esomeprazole capsules to allow completion of the study. The same lot number will be used throughout the study.

The lot numbers and expiration dates (where available) of the study drugs supplied will be recorded in the final report.

Records will be made of the receipt, preparation, dispensing, and final disposition of the study drugs supplied. All study drugs will be prepared and labeled by licensed pharmacy staff according to the procedures outlined in the pharmacy manual.

### 8.1.5 Clinical Study Drug Blinding

This is an open-label study.

## 8.1.6 Randomization Code Creation and Storage

NA

### 8.1.7 Clinical Trial Blind Maintenance/Unblinding Procedure

NA

### Accountability and Destruction of Sponsor-Supplied Drugs 8.1.8

licable reims of Use At the conclusion of the study, any unused TAK-906 and esomeprazole study drug will be retained by Celerion, returned to the Sponsor or designee, or destroyed, as per Sponsor instructions. If no supplies remain, this fact will be documented in the pharmacy product accountability records.

er Sponduct acc adults only and subject to state only and subject to s

### 9.0 STUDY PROCEDURES

### 9.1 Administrative Procedures

### 9.1.1 Informed Consent Procedure

The purpose of the study, the procedures to be carried out and the potential hazards will be described to the subjects in non-technical terms. Subjects will be required to read, sign, and date an ICF summarizing the discussion prior to screening, and will be assured that they may withdraw from the study at any time without jeopardizing their medical care.

Subjects will be given a copy of their signed ICF.

### 9.1.1.1 Assignment of Screening and Randomization Numbers

Each subject will be assigned a unique identification number upon screening. Subjects who complete the study screening assessments and meet all the eligibility criteria will be assigned a unique identification number at the time of the first dosing, different from the screening number.

If replacement subjects are used, the replacement subject number will be 100 more than the original (eg, Subject No. 101 will replace Subject No. 1).

## 9.1.1.2 Study Drug Assignment

This is a fixed-sequence (1-way crossover) study. All subjects will receive the same treatments as detailed in Section 6.1.

### 9.1.2 Inclusion and Exclusion

### 9.1.2.1 Inclusion Criteria

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

- 1. Healthy, adult, male or female, 18-55 years of age, inclusive, at screening.
- 2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study, based on screening urine cotinine test.
- 3. Body mass index (BMI)  $\geq$ 18.0 and  $\leq$ 30.0 kg/m<sup>2</sup> at screening.
- 4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the principal Investigator or designee.
- 5. For a male or female of non-childbearing potential, use acceptable birth control methods as indicated in Appendix D.
- 6. A male subject who is nonsterilized and sexually active with a female partner of childbearing potential must agree to use a barrier method of contraception from signing of the ICF throughout the duration of the study and through to the follow up (ie, 10-14 days after the last dose of TAK-906) (refer to Appendix D).

- 7. If male, must agree not to donate sperm from the first dosing until follow-up visit (10-14 days after the last dosing).
- 8. Understands the study procedures in the ICF, and be willing and able to comply with the protocol.

### 9.1.2.2 Exclusion Criteria

The subject must be excluded from participating in the study if the subject:

- 1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
- 2. History or presence of clinically significant endocrine, gastrointestinal (including motility disorder and intestinal obstruction), cardiovascular, hematological, hepatic, immunological, renal, respiration, genitourinary, or major neurological (including stroke and chronic seizures) any other clinically significant abnormalities or disease in the opinion of the Investigator or designee.
- 3. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
- 4. History of cancer (malignancy).
- 5. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
- 6. History or presence of hypersensitivity or idiosyncratic reaction to TAK-906 or related compounds, or to esomeprazole or PPIs (see NEXIUM® USPI).
- 7. Female subjects of childbearing potential.
- 8. Female subjects with a positive pregnancy test or who is lactating.
- 9. Positive urine drug or alcohol results at screening or first check-in.
- 10. Positive urine cotinine at screening.
- 11. Positive results at screening for HIV, HBsAg, or HCV.
- 12. QTcF interval is >450 msec or ECG findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
- 13. Estimated creatinine clearance <90 mL/min at screening.
- 14. Unable to refrain from or anticipates the use of:
  - Any drug, including prescription and non-prescription medications (including PPIs, antacids, and H<sub>2</sub>-antagonist), herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Thyroid hormone replacement medication may be permitted if the subject has been on the same stable dose for the immediate 3 months prior to first study drug administration. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the Investigator or designee.

- Any drugs known to significantly affect the absorption, distribution, metabolism, or elimination of study drugs (TAK-906 or esomeprazole) within 28 days prior to the first dosing and throughout the study. Appropriate sources (eg, Flockhart Table<sup>TM</sup>) will be consulted to confirm lack of PK/pharmacodynamic interaction with study drug.
- 15. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
- 16. Donation of blood or significant blood loss (eg, approximately 500 mL) within 56 days prior to the first dosing.
- 17. Plasma donation within 7 days prior to the first dosing.
- 18. Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Study Period 1 of the current study.

## 9.1.3 Medical History/Demography

Medical history and demographic data, including name, sex, age, race, ethnicity, and history of tobacco use will be recorded.

### 9.1.4 Concomitant Medications

Concomitant medications will be prohibited as listed in Section 7.1 and in Section 9.1.2.2. All medications taken by subjects during the course of the study will be recorded.

## 9.2 Clinical Procedures and Assessments

The Schedule of Study Procedures (Section 3.0) summarizes the clinical procedures to be performed at each visit. Individual clinical procedures are described in detail below. Additional evaluations/testing may be deemed necessary by the Investigator or designee and/or the Sponsor for reasons related to subject safety.

For this study, the collection of blood for plasma TAK-906 concentrations is the critical parameter and samples need to be collected as close to the exact time point as possible. All other procedures should be completed as close to the prescribed/scheduled time as possible, but can be performed prior or after the prescribed/scheduled time.

Any nonscheduled procedures required for urgent evaluation of safety concerns take precedence over all routine scheduled procedures.

### 9.2.1 Full Physical Exam

A full physical examination will be performed as outlined in the Schedule of Study Procedures (Section 3.0). Symptom-driven physical examinations may be performed at other times, if deemed necessary by the Investigator or designee.

### 9.2.2 Height and Weight

icable reinsofus Body height (cm) and weight (kg) will be reported as outlined in the Schedule of Study Procedures (Section 3.0).

### 9.2.3 **BMI**

BMI will be calculated based on the height and weight measured at screening.

### 9.2.4 Vital Signs

Single measurements of body temperature, respiratory rate, blood pressure and heart rate, will be measured as outlined in the Schedule of Study Procedures (Section 3.0). Additional vital signs may be taken at any other times, if deemed necessary.

Blood pressure and heart rate measurements will be performed with subjects in a supine position, except when they are supine or semi-recumbent because of study procedures and/or AEs (eg., nausea, dizziness) or if deemed necessary by the Investigator or designee. Subjects should have rested in a supine position for at least 5 minutes before the measurements.

Blood pressure and heart rate will be measured within 24 hours prior to Day 1 dosing of each treatment period for the predose time point. When scheduled postdose, vital signs will be performed within approximately 15 minutes of the scheduled time point.

### 9.2.5 12-Lead ECG

Single 12-lead ECGs will be performed as outlined in the Schedule of Study Procedures (Section 3.0). Additional ECGs may be taken at any other times, if deemed necessary by the investigator or designee.

ECGs will be performed with subjects in a supine position and subjects should have rested in a supine position for at least 5 minutes before recording the ECG. All ECG tracings will be reviewed by the investigator or designee.

ECGs will be measured within 24 hours prior to Day 1 dosing of each period for the predose time point. When scheduled postdose, ECGs will be performed within approximately 20 minutes of the scheduled time point.

### 9.2.6 Study Drug Administration

TAK-906 oral capsule and esomeprazole oral capsule will be provided as described in Section 8.1.

Subjects will be instructed not to crush, split, or chew the TAK-906 or esomeprazole capsules. Capsules should be swallowed as whole.

Treatments A and B are described as:

25 mg TAK-906 (1 x 25 mg TAK-906 capsule) Study Period 1 (Treatment A):

40 mg esomeprazole (1 x 40 mg Nexium® capsule, or Study Period 2 (Treatment B):

generic equivalent) QD for 5 days (Days 1 through 5 of

Study Period 2) with 25 mg TAK-906 (1 x 25 mg TAK-906 capsule) administered 1 hour following esomeprazole dose on Day 4 of Study Period 2.

The oral doses of TAK-906 will be administered following an overnight fast with approximately 240 mL of water. The oral doses of esomeprazole on Days 1 to 3 and 5 of Study Period 2 will be administered following a fast of at least 2 hours.

The exact clock time of oral dosing will be recorded.

### 9.2.7 AE Monitoring

Subjects will be monitored throughout the study for AEs to the study formulations and/or procedures as described in Section 10.0.

## 9.2.8 Laboratory Procedures and Assessments

All tests listed below will be performed as outlined in the Schedule of Study Procedures (Section 3.0). In addition, laboratory safety tests may be performed at various unscheduled time points, if deemed necessary by the Investigator or designee.

### 9.2.9 Clinical Laboratory Tests

### <u>Hematology</u>

Hematology will consist of the following tests:

| Hemoglobin | Red blood cell count |
|----------------------------------------|----------------------|
| Hematocrit | Platelet count |
| Total and differential leukocyte count | |

### Chemistry

Serum chemistry tests will be performed after at least an 8-hour fast; however, in case of dropouts or rechecks, subjects may not have fasted for 8 hours prior to the serum chemistry sample being taken.

Chemistry evaluations will consist of the following standard chemistry panel:

| Total protein | Albumin |
|----------------------------------|--------------|
| Blood Urea Nitrogen | Sodium |
| Bilirubin (total and direct) | Potassium |
| Alkaline phosphatase | Chloride |
| Aspartate aminotransferase (AST) | Glucose |
| Alanine aminotransferase (ALT) | Creatinine * |

<sup>\*</sup> At screening, creatinine clearance will be calculated using the Cockcroft-Gault formula.

### Urinalysis

Urinalysis will consist of the following tests:

| рН | Bilirubin | 101 |
|------------------|----------------------|-------|
| Specific gravity | Blood * | |
| Protein * | Nitrite * | |
| Glucose | Urobilinogen | . ( . |
| Ketones | Leukocyte esterase * | · |

<sup>\*</sup> If urinalysis is positive for protein, blood, nitrite and/or leukocyte esterase, a microscopic examination (for red blood cells, white blood cells, bacteria, casts, and epithelial cells) will be performed.

### Other

| Urine drug screen |
|---|
| Opiates (includes morphine, heroin (diacetylmorphine), |
| codeine, 6-acetylmorphine, dihydrocodeine, hydrocodone, thebaine, and, hydromorphone) |
| — Amphetamines |
| _ Barbiturates |
| Benzodiazepines |
| Cocaine |
| Cannabinoids |

9.3 PK SamplesPrimary specimen collection parameters are provided in Table 9.a.

For all subjects, blood samples for the determination of plasma TAK-906 will be collected at scheduled time points as delineated in the Schedule of Study Procedures (Section 3.0) in 4 mL blood collection tubes containing the appropriate anticoagulant, respectively. The actual time of sample collection will be recorded on the source document in the case report form (CRF).

Instruction for blood sampling, collection, processing, and sample shipment will be provided separately.

| Table 9.a | <b>Primary</b> | Specimen | Collections |
|-----------|----------------|----------|-------------|
|-----------|----------------|----------|-------------|

| Study ID TAK-906-1006 | | | | Page 33 of 68 |
|---|---|---|---|---|
| Protocol Final | | | | 04 Feb 2019 |
| Table 9.a Primary S <sub>I</sub> | oecimen Collec | etions | | |
| | | Primary | | ~~ |
| | Primary | Specimen | | Sample |
| Specimen Name | Specimen | Derivative | <b>Description of Intended Use</b> | Collection |
| Plasma sample for PK | Plasma | | PK analysis | Mandatory |
| CCI | | | | |

### 9.3.1 **PK Measurements**

### 9.3.2 **PK Measurements**

### 9.3.2.1 Plasma PK Measurements

ine applic The PK parameters of TAK-906 will be derived using noncompartmental analysis methods and will be determined from the concentration-time data for all evaluable subjects. Actual sampling times, rather than scheduled sampling times, will be used in all PK computations involving sampling times. A more detailed description will be given in the clinical pharmacology analysis plan.

PK parameters for plasma TAK-906 and concentrations will be calculated as follows, as appropriate, following oral administration:

The area under the concentration-time curve from time 0 to time of the last quantifiable AUC<sub>last</sub>:

concentration.

AUCinf: Area under the concentration-time curve from time 0 to infinity, calculated using the

observed value of the last quantifiable concentration.

Maximum observed concentration.



Other PK parameters may be calculated if deemed necessary for the interpretation of the data. All efforts will be made to obtain the PK samples at the exact nominal time relative to dosing. However, samples obtained within 10% of the nominal time from dosing will not be captured as a protocol deviation, as long as the exact time of the sample collection is noted on CRF.

The decision as to which plasma samples collected will be assayed for evaluation of PK will be determined by the sponsor. If indicated, these samples may also be assayed and/or pooled for assay in an exploratory manner for metabolites.



### 9.3.4 Confinement

In Study Period 1, subjects will be housed on Day -1, at the time indicated by the CRU until after the 48-hour blood draw and/or study procedures on Day 3. In Study Period 2, Subjects will be housed on Day 3 at the time indicated by the CRU until after the 48-hour blood draw and/or study procedures on Day 6.

Subjects will return for dosing and/or study procedures as indicated in the Schedule of Study Procedures (Section 3.0). A subject may be required to remain at the CRU for longer at the discretion of the Investigator or designee.

As per site preference, subjects may be confined throughout the washout period.

Property of Takedai. For non-corr

An AE is defined as any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study; it does not necessarily have to have a causal relationship with the treatment.

An AE can therefore be any unfavorable laboratory for the study of the study

laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.

An untoward finding generally may:

- Indicate a new diagnosis or unexpected worsening of a preexisting condition. (Intermittent events for pre-existing conditions or underlying disease should not be considered AEs.)
- Necessitate therapeutic intervention.
- Require an invasive diagnostic procedure.
- Require discontinuation or a change in dose of study medication or a concomitant medication.
- Be considered unfavorable by the investigator for any reason.

Diagnoses versus signs and symptoms:

Each event should be recorded to represent a single diagnosis. Accompanying signs (including abnormal laboratory values or ECG findings) or symptoms should NOT be recorded as additional AEs. If a diagnosis is unknown, sign(s) or symptom(s) should be recorded appropriately as an AE(s).

Laboratory values and ECG findings:

- Changes in laboratory values or ECG parameters maybe considered AEs if they are judged to be clinically significant (ie, if some action or intervention is required or if the investigator judges the change to be beyond the range of normal physiologic fluctuation). A laboratory re-test and/or continued monitoring of an abnormal value are not considered an intervention. In addition, repeated or additional noninvasive testing for verification, evaluation or monitoring of an abnormality is not considered an intervention.
- If abnormal laboratory values or ECG findings are the result of pathology for which there is an overall diagnosis (eg, increased creatinine in renal failure), the diagnosis only should be reported appropriately as an AE.

Pre-existing conditions:

A pre-existing condition (present at the time of signing of informed consent) is considered a concurrent medical history condition and should NOT be recorded as an AE. A baseline evaluation (eg, laboratory test, ECG, X-ray, etc) should NOT be recorded as an AE unless related to a study procedure. However, if the subject experiences a worsening or complication
of such a concurrent medical history condition, the worsening or complication should be recorded appropriately as an AE (worsening or complication occurs after informed consent is signed). Investigators should ensure that the event term recorded captures the change in the condition (eg, "worsening of...").

- If a subject has a pre-existing episodic condition (eg, asthma, epilepsy), any occurrence of an episode should only be captured as an AE if the episodes become more frequent, serious, or severe in nature, that is, investigators should ensure that the AE term recorded captures the change from Baseline in the condition (eg "worsening of...").
- If a subject has a degenerative concurrent condition (eg, cataracts, rheumatoid arthritis), worsening of the condition should only be captured as an AE if occurring to a greater extent to that which would be expected. Again, investigators should ensure that the AE term recorded captures the change in the condition (eg, "worsening of...").

### Worsening of AEs:

• If the subject experiences a worsening or complication of an AE after the first administration of study medication or after any change in study medication, the worsening or complication should be recorded as a new AE. Investigators should ensure that the AE term recorded captures the change in the condition (eg, "worsening of...").

### Changes in severity of AEs:

• If the subject experiences a change in the severity of an AE that is not associated with a change in study medication, the event should be captured once with the maximum severity recorded.

# Preplanned surgeries or procedures:

Preplanned procedures (surgeries or therapies) that were scheduled prior to signing of
informed consent are not considered AEs. However, if a preplanned procedure is performed
early (eg, as an emergency) due to a worsening of the pre-existing condition, the worsening of
the condition should be captured appropriately as an AE. Complications resulting from any
planned surgery should be reported as AEs.

# Elective surgeries or procedures:

• Elective procedures performed where there is no change in the subject's medical condition should not be recorded as AEs but should be documented in the subject's source documents. Complications resulting from an elective surgery should be reported as AEs.

### Overdose:

- An overdose is defined as a known deliberate or accidental administration of investigational drug, to or by a study subject, at a dose above that which is assigned to that individual subject according to the study protocol. It is up to the investigator or the reporting physician to decide whether a dose is to be considered an overdose, in consultation with the Sponsor.
- All cases of overdose (with or without associated AEs) will be documented on an Overdose page of the (e)CRF, in order to capture this important safety information consistently in the

database. AEs associated with an overdose will be documented on AE CRF(s) according to Section 10.0.

- Serious adverse events (SAEs) of overdose should be reported according to the procedure outlined in Section 10.2.8.
- In the event of drug overdose, the subject should be treated symptomatically.

### 10.1.1 SAEs

An SAE is defined as any untoward medical occurrence that at any dose:

- 1. Results in DEATH.
- 2. Is LIFE THREATENING.
  - The term "life threatening" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.
- 3. Requires inpatient HOSPITALIZATION or prolongation of existing hospitalization.
- 4. Results in persistent or significant DISABILITY/INCAPACITY.
- 5. Is a CONGENITAL ANOMALY/BIRTH DEFECT.
- 6. Is an IMPORTANT MEDICAL EVENT assessed by the Investigator and/or the Sponsor, that satisfies any of the following:
  - May require intervention to prevent items 1 through 5 above.
  - May expose the subject to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.
- Includes any event of synonym described in the Takeda Medically Significant AE List (Table 10.a).

  Productive of the Takeda Medically Significant AE List (Table 10.a).

**Table 10.a** Takeda Medically Significant AE List

| Term | |
|---|---|
| Acute respiratory failure/acute respiratory | Hepatic necrosis |
| distress syndrome | Acute liver failure |
| Torsade de pointes / ventricular fibrillation / | Anaphylactic shock |
| ventricular tachycardia | Acute renal failure |
| Malignant hypertension | Pulmonary hypertension |
| Convulsive seizures | Pulmonary fibrosis |
| Agranulocytosis | Confirmed or suspected endotoxin shock |
| Aplastic anemia | Confirmed or suspected transmission of infectious agent by |
| Toxic epidermal necrolysis/ | a medicinal product |
| Stevens-Johnson syndrome | Neuroleptic malignant syndrome / malignant hyperthermia |
| | Spontaneous abortion / stillbirth and fetal death |

AEs that fulfill 1 or more of the serious criteria above are to be considered SAEs and should be reported and followed up in the same manner (see Sections 10.1 and 10.1.1).

### 10.1.2 Special Interest AEs

NA

### 10.2 AE Procedures

# 10.2.1 Assigning Severity/Intensity of AEs

The PI or designee will review each AE and assess its relationship to drug treatment (refer to Section 10.2.2). All AEs, including signs, symptoms, or clinically significant treatment-emergent laboratory abnormalities will be graded on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 toxicity grading scale.

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on the following general guideline [9]:

| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
|---|---|
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL*. |
| Grade 3 | Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL**. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE. |

A Semi-colon indicates 'or' within the description of the grade.

Note: Not all grades are appropriate for all AEs. Therefore, some AEs are listed within the CTCAE with fewer than 5 options for grade selection. Grade 5 (death) is not appropriate for some AEs and therefore is not an option. ADL=Activities of Daily Living

### 10.2.2 Assigning Causality of AEs

The relationship of each AE to study medication(s) will be assessed using the following categories:

Related:

An AE that follows a reasonable temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which a causal relationship is at least a reasonable possibility, ie, the relationship cannot be ruled out, although factors other than the drug, such as underlying diseases, complications, concomitant drugs and concurrent treatments, may also be responsible.

Not Related:

An AE that does not follow a reasonable temporal sequence from administration of a drug and/or that can reasonably be explained by other factors, such as underlying diseases, complications, concomitant medications and concurrent treatments.

### 10.2.3 Start Date

The start date of the AE is the date that the first signs/symptoms were noted by the subject and/or investigator.

<sup>\*</sup> Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

<sup>\*\*</sup> Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

### **10.2.4 End Date**

The end date of the AE is the date at which the subject recovered, the event resolved but with sequelae or the subject died.

### **10.2.5** Pattern of Adverse Event (Frequency)

Episodic AEs (eg, headache) or those which occur repeatedly over a period of consecutive days are intermittent. All other events are continuous.

### 10.2.6 Action Taken With Study Treatment

- Drug withdrawn a study medication is stopped due to the particular AE.
- Dose not changed the particular AE did not require stopping a study medication.
- Unknown only to be used if it has not been possible to determine what action has been taken.
- Not applicable a study medication was stopped for a reason other than the particular AE eg, the study has been terminated, the subject died, dosing with study medication had not yet started or dosing with study medication was already stopped before the onset of the AE.
- Dose reduced the dose was reduced due to the particular AE.
- Dose increased the dose was increased due to the particular AE.
- Drug interrupted the dose was interrupted due to the particular AE.

### **10.2.7 Outcome**

- Recovered/resolved subject returned to first assessment status with respect to the AE.
- Recovering/resolving the intensity is lowered by one or more stages: the diagnosis has or signs/symptoms have almost disappeared; the abnormal laboratory value improved, but has not returned to the normal range or to the baseline value; the subject died from a cause other than the particular AE with the condition remaining "recovering/resolving."
- Not recovered/not resolved there is no change in the diagnosis, signs or symptoms; the intensity of the diagnosis, signs/symptoms or laboratory value on the last day of the observed study period has become worse than when it started; is an irreversible congenital anomaly; the subject died from another cause with the particular AE state remaining "Not recovered/not resolved."
- Recovered/ Resolved with sequelae the subject recovered from an acute AE but was left with permanent/significant impairment (eg, recovered from a cardiovascular accident but with some persisting paresis).
- Fatal an AE that is considered as the cause of death.
- Unknown the course of the AE cannot be followed up due to hospital change or residence change at the end of the subject's participation in the study.

Collection of AEs (ie, AEs, SAEs, Special Interest AEs, and Abnormal LFTs) will commence at the time the subject signs the informed consent. Routine collection of AEs will continue until a follow-up visit on Day 10-14 after the last dose of TAK-906 For subthe administration of study medication. participation.

### 10.2.8.2 Reporting AEs

At each study visit, the investigator will assess whether any subjective AEs have occurred. A neutral question, such as "How have you been feeling since your last visit?" may be asked. Subjects may report AEs occurring at any other time during the study. Subjects experiencing an SAE prior to the first exposure to investigational product must be monitored until the symptoms subside and any clinically relevant changes in laboratory values have returned to Baseline or there is a satisfactory explanation for the change. Nonserious AEs that begin prior to the first exposure to investigational product, related or unrelated to the study procedure, need not be followed-up for the purposes of the protocol.

All subjects experiencing AEs, whether considered associated with the use of the study medication or not, must be monitored until the symptoms subside and any clinically relevant changes in laboratory values have returned to Baseline or until there is a satisfactory explanation for the changes observed. All AEs will be documented in the AE page of the CRF, whether or not the investigator concludes that the event is related to the drug treatment. The following information will be documented for each event:

- Event term.
- Start and end date and time.
- Pattern of AE (frequency).
- Severity/Intensity.
- Causality (Investigator's opinion of the causal relationship between the event and administration of study drug[s]).
- Action taken with study drug.
- Outcome of event.
- Seriousness.

### 10.2.8.3 Reporting SAEs

When an SAE occurs through the AE collection period it should be reported according to the procedure outlined below:

A Takeda SAE form must be completed, in English and signed by the investigator immediately or within 24 hours of first onset or notification of the event. The information should be completed as fully as possible but contain, at a minimum:

- A short description of the event and the reason why the event is categorized as serious.
- Subject identification number.
- Investigator's name.
- Name of the study medication(s).
- Causality assessment.

The SAE form should be transmitted within 24 hours to the attention of the contact listed in Section 14.1.1.

Any SAE spontaneously reported to the investigator following the AE collection period should be reported to the Sponsor if considered related to study participation.

Reporting of SAEs that begin before first administration of investigational product will follow the same procedure for SAEs occurring on treatment.

### SAE Follow-Up

If information is not available at the time of the first report becomes available at a later date, the investigator should complete a follow-up SAE form or provide other written documentation and fax it immediately within 24 hours of receipt. Copies of any relevant data from the hospital notes (eg, ECGs, laboratory tests, discharge summary, postmortem results) should be sent to the addressee, if requested.

All SAEs should be followed up until resolution or permanent outcome of the event. The timelines and procedure for follow-up reports are the same as those for the initial report.

10.2.8.4 Reporting Special Interest AEs

NA

### 10.2.8.5 Reporting of Abnormal LFTs

If a subject is noted to have ALT or AST elevated >3 ×ULN on 2 consecutive occasions, the abnormality should be recorded as an AE. In addition, an LFT Increases CRF must be completed providing additional information on relevant recent history, risk factors, clinical signs and symptoms and results of any additional diagnostic tests performed.

If a subject is noted to have ALT or AST >3 ×ULN and total bilirubin >2 ×ULN for which an alternative etiology has not been identified, the event should be recorded as an SAE and reported as per Section 10.2.8.3. The investigator must contact the Medical Monitor for discussion of the relevant subject details and possible alternative etiologies, such as acute viral hepatitis A or B or other acute liver disease. Follow-up laboratory tests as described in Section 9.2.8 must also be

performed. In addition, an LFT Increases CRF must be completed and transmitted with the Takeda SAE form (as per Section 10.2.9).

### 10.2.9 Safety Reporting to Investigators, IRBs or IECs, and Regulatory Authorities

The Sponsor will be responsible for reporting all suspected unexpected serious adverse reactions (SUSARs) and any other applicable SAEs to regulatory authorities, investigators and IRBs or IECs, as applicable, in accordance with national regulations in the countries where the study is conducted. Relative to the first awareness of the event by/or further provision to the Sponsor or Sponsor's designee, SUSARs will be submitted within 7 days for fatal and life-threatening events and 15 days for other serious events, unless otherwise required by national regulations. The Sponsor will also prepare an expedited report for other safety issues where these might materially alter the current benefit-risk assessment of an investigational medicinal product or that would be  and se sufficient to consider changes in the investigational medicinal products administration or in the overall conduct of the study. The investigational site also will forward a copy of all expedited reports to his or her IRB or IEC in accordance with national regulations.

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a SAP. The SAP will be prepared by Celerion and agreed upon with the Sponsor. This document may modify the plans outlined in the protocol. I modifications of the primary endpoints definition protocol amendment. A Jan. be performed if deemed appropriate. to the of

### 11.1.1 Analysis Sets

11.1.1.1 Safety Set

All subjects who received at least one dose of the study drug will be included in the safety evaluations.

11.1.1.2 PK Set

Samples from all subjects will be assayed even if the subjects do not complete the study. All subjects who comply sufficiently with the protocol and display an evaluable PK profile (eg, exposure to treatment, availability of measurements and absence of major protocol violations) will be included in the statistical analyses.

11.1.1.3 PD Set

NA

# 11.1.2 Analysis of Demography and Other Baseline Characteristics

Continuous demographic data (ie, age, weight, height, and BMI) will be listed and summarized using appropriate summary statistics. Categorical demographic data (ie, gender, race, and ethnicity) will also be listed and tabulated.

### 11.1.3 PK Analysis

Descriptive statistics will be provided for the plasma TAK-906 concentrations using appropriate summary statistics to be fully specified in the SAP.

PK parameters for plasma TAK-906 concentrations will be calculated as described in Section 9.3.2.1.

For evaluation of potential effect of esomeprazole on TAK-906 PK, an ANOVA will be performed on the In-transformed C<sub>max</sub>, AUC<sub>last</sub>, and AUC<sub>inf</sub>. The ANOVA model will include treatment as

fixed effect and subject as a random effect. Each ANOVA will include calculation of least-squares means (LSM) as well as the difference between treatment LSM. The geometric mean of the relative bioavailability of the TAK-906 with esomeprazole regimen relative to the TAK-906 regimen alone and the associated 90% CIs will be determined by exponentiation of the appropriate estimates for the difference between regimens in the log-transformed parameters

### 11.1.4 PD Analysis

NA

### 11.1.5 Safety Analysis

All safety data will be populated in the individual CRFs.

Dosing dates and times will be listed by subject.

Quantitative safety data as well as the difference to baseline, when appropriate, will be summarized using the appropriate descriptive statistics.

### 11.1.5.1 AEs

AEs will be coded using the most current version of Medical Dictionary for Regulatory Activities (MedDRA®) available at Celerion and summarized by treatment for the number and percentage of subjects reporting the TEAE and the number of TEAEs reported. A by-subject AE data listing including verbatim term, coded term, treatment, severity, and relationship to treatment will be provided.

### 11.1.5.2 Clinical Laboratory Evaluation

Clinical laboratory results will be summarized by treatment and point of time of collection and a shift table describing out of normal range shifts will be provided.

### 11.1.5.3 Vital Signs and ECG Parameters

Vital signs and ECG assessments will be summarized by treatment and point of time of collection.

### 11.1.5.4 Physical Examination

Physical examination findings will be presented in the data listings.

# 11.2 Interim Analysis and Criteria for Early Termination

No interim analysis is planned.

### 11.3 Determination of Sample Size

The total of twelve (12) subjects will be enrolled in this study. This sample size will provide at least 80% power to conclude the  $C_{max}$  of TAK-906 will not decrease more than 50% in the presence of esomeprazole, assuming that the intra-subject %CV for  $C_{max}$  of TAK-906 will not

exceed 45% and a true ratio of 0.8. Lower intra-subject variability was observed for AUC in previous studies; therefore, the power is expected to be greater for AUC.

 and subject to the applic

Monitoring visits to the study site will be made periodically during the study to ensure that all aspects of the protocol are followed. Source documents will be reviewed for verification of dark recorded on the CRFs. Source documents are defined as original document.

The investigator and study site guarantee access to designee (Contract Research Contract Research Contr

All aspects of the study and its documentation will be subject to review by the Sponsor or the Sponsor's designee (as long as blinding is not jeopardized), including but not limited to the Investigator's Binder, study drug, subject medical records, informed consent documentation, and review of CRFs and associated source documents. It is important that the investigator and other study personnel are available during the monitoring visits and that sufficient time is devoted to the process.

### 12.2 **Protocol Deviations**

The investigator should not deviate from the protocol, except where necessary to eliminate an immediate hazard to study subjects. Should other unexpected circumstances arise that will require deviation from protocol-specified procedures, the investigator should consult with the sponsor or designee (and IRB or IEC, as required) to determine the appropriate course of action. There will be no exemptions (a prospectively approved deviation) from the inclusion or exclusion criteria.

Significant deviations include, but are not limited to, those that involve fraud or misconduct, increase the health risk to the subject, or confound interpretation of primary study assessment.

### **Quality Assurance Audits and Regulatory Agency Inspections** 12.3

The study site also may be subject to quality assurance audits by the Sponsor or designees. In this circumstance, the Sponsor-designated auditor will contact the site in advance to arrange an auditing visit. The auditor may ask to visit the facilities where laboratory samples are collected, where the medication is stored and prepared, and any other facility used during the study. In addition, there is the possibility that this study may be inspected by regulatory agencies, including those of foreign governments (eg, the FDA, the United Kingdom Medicines and Healthcare products Regulatory Agency, the Pharmaceuticals and Medical Devices Agency of Japan). If the study site is contacted for an inspection by a regulatory body, the Sponsor should be notified immediately. The investigator guarantees access for quality assurance auditors to all study documents as described in Section 12.1.

### 13.0 ETHICAL ASPECTS OF THE STUDY

This study will be conducted with the highest respect for the individual participants (ie, subjects) according to the protocol, the ethical principles that have their origin in the Declaration of Helsinki, and the International Council for Harminsation (ICH) Harmonised Tripartite Guideline for GCP. Each investigator will conduct the study according to applicable local or regional regulatory requirements and align his or her conduct in accordance with the "Responsibilities of the Investigator" that are listed in Appendix A. The principles of Helsinki are addressed through the protocol and through appendices containing requirements for informed consent and investigator responsibilities.

### 13.1 IRB and/or IEC Approval

IRBs and IECs must be constituted according to the applicable state and federal/local requirements of each participating region. The Sponsor or designee will require documentation noting all names and titles of members who make up the respective IRB or IEC. If any member of the IRB or IEC has direct participation in this study, written notification regarding his or her abstinence from voting must also be obtained. Those Americas sites unwilling to provide names and titles of all members due to privacy and conflict of interest concerns should instead provide a Federal Wide Assurance Number or comparable number assigned by the Department of Health and Human Services.

The Sponsor or designee will supply relevant documents for submission to the respective IRB or IEC for the protocol's review and approval. This protocol, the Investigator's Brochure, a copy of the ICF, and, if applicable, subject recruitment materials and/or advertisements and other documents required by all applicable laws and regulations, must be submitted to a central or local IRB or IEC for approval. The IRB's or IEC's written approval of the protocol and subject informed consent must be obtained and submitted to the Sponsor or designee before commencement of the study (ie, before shipment of the Sponsor-supplied drug or study specific screening activity). The IRB or IEC approval must refer to the study by exact protocol title, number, and version date; identify versions of other documents (eg, ICF) reviewed; and state the approval date. The Sponsor will ship drug/notify site once the Sponsor has confirmed the adequacy of site regulatory documentation and, when applicable, the Sponsor has received permission from competent authority to begin the study. Until the site receives drug/notification no protocol activities, including screening, may occur.

Sites must adhere to all requirements stipulated by their respective IRB or IEC. This may include notification to the IRB or IEC regarding protocol amendments, updates to the ICF, recruitment materials intended for viewing by subjects, local safety reporting requirements, reports and updates regarding the ongoing review of the study at intervals specified by the respective IRB or IEC, and submission of the investigator's final status report to IRB or IEC. All IRB and IEC approvals and relevant documentation for these items must be provided to the Sponsor or its designee.

Subject incentives should not exert undue influence for participation. Payments to subjects must be approved by the IRB or IEC and Sponsor.

### Subject Information, Informed Consent, and Subject Authorization 13.2

ins of Use Written consent documents will embody the elements of informed consent as described in the Declaration of Helsinki and the ICH Guidelines for GCP and will be in accordance with all applicable laws and regulations. The ICF, subject authorization form (if applicable), and subject information sheet (if applicable) describe the planned and permitted uses, transfers, and disclosures of the subject's personal and personal health information for purposes of conducting the study. The ICF and the subject information sheet (if applicable) further explain the nature of the study, its objectives, and potential risks and benefits, as well as the date informed consent is given. The ICF will detail the requirements of the participant and the fact that he or she is free to withdraw at any time without giving a reason and without prejudice to his or her further medical care.

The investigator is responsible for the preparation, content, and IRB or IEC approval of the ICF and, if applicable, the subject authorization form. The ICF, subject authorization form (if applicable), and subject information sheet (if applicable) must be approved by both the IRB or IEC and the Sponsor prior to use.

The ICF, subject authorization form (if applicable), and subject information sheet (if applicable) must be written in a language fully comprehensible to the prospective subject. It is the responsibility of the investigator to explain the detailed elements of the ICF, subject authorization form (if applicable), and subject information sheet (if applicable) to the subject. Information should be given in both oral and written form whenever possible and in the manner deemed appropriate by the IRB or IEC. In the event the subject is not capable of rendering adequate written informed consent, then the subject's legally acceptable representative may provide such consent for the subject in accordance with applicable laws and regulations.

The subject, or the subject's legally acceptable representative, must be given ample opportunity to: (1) inquire about details of the study, and (2) decide whether or not to participate in the study. If the subject, or the subject's legally acceptable representative, determines he or she will participate in the study, then the ICF and subject authorization form (if applicable) must be signed and dated by the subject, or the subject's legally acceptable representative, at the time of consent and prior to the subject entering into the study. The subject or the subject's legally acceptable representative should be instructed to sign using their legal names, not nicknames, using blue or black ballpoint ink. The investigator must also sign and date the ICF and subject authorization (if applicable) at the time of consent and prior to subject entering into the study; however, the Sponsor may allow a designee of the investigator to sign to the extent permitted by applicable law.

Once signed, the original ICF, subject authorization form (if applicable), and subject information sheet (if applicable) will be stored in the investigator's site file. The investigator must document the date the subject signs the informed consent in the subject's medical record. Copies of the signed ICF, the signed subject authorization form (if applicable), and subject information sheet (if applicable) shall be given to the subject.

All revised ICFs must be reviewed and signed by relevant subjects or the relevant subject's legally acceptable representative in the same manner as the original informed consent. The date the

subjects who consented and provided a blood sample for DNA analysis can withdraw their consent and request disposal of a stored sample at any time prior to analysis. Notify Sponsor of consent withdrawal.

13.3 Subject Confidentiality

The Sponsor and designs

against invasion of privacy. Throughout this study, a subject's source data will only be linked to the Sponsor's clinical study database or documentation via a unique identification number. As permitted by all applicable laws and regulations, limited subject attributes, such as sex, age, or date of birth, and subject initials may be used to verify the subject and accuracy of the subject's unique identification number.

To comply with ICH Guidelines for GCP and to verify compliance with this protocol, the Sponsor requires the investigator to permit its monitor or designee's monitor, representatives from any regulatory authority (eg, FDA, Medicines and Healthcare products Regulatory Agency, Pharmaceuticals and Medical Devices Agency), the Sponsor's designated auditors, and the appropriate IRBs and IECs to review the subject's original medical records (source data or documents), including, but not limited to, laboratory test result reports, ECG reports, admission and discharge summaries for hospital admissions occurring during a subject's study participation, and autopsy reports. Access to a subject's original medical records requires the specific authorization of the subject as part of the informed consent process (see Section 13.2).

Copies of any subject source documents that are provided to the Sponsor must have certain personally identifiable information removed (ie, subject name, address, and other identifier fields not collected on the subject's CRF).

### Publication, Disclosure, and Clinical Trial Registration Policy 13.4

### 13.4.1 Publication and Disclosure

The investigator is obliged to provide the Sponsor with complete test results and all data derived by the investigator from the study. During and after the study, only the Sponsor may make study information available to other study investigators or to regulatory agencies, except as required by law or regulation. Except as otherwise allowable in the clinical study site agreement, any public disclosure (including publicly accessible websites) related to the protocol or study results, other than study recruitment materials and/or advertisements, is the sole responsibility of the Sponsor.

The Sponsor may publish any data and information from the study (including data and information generated by the investigator) without the consent of the investigator. Manuscript authorship for any peer-reviewed publication will appropriately reflect contributions to the production and review of the document. All publications and presentations must be prepared in accordance with this section and the Clinical Study Site Agreement. In the event of any discrepancy between the protocol and the Clinical Study Site Agreement, the Clinical Study Site Agreement will prevail.

### 13.4.2 Clinical Trial Registration

In order to ensure that information on clinical studies reaches the public in a timely manner and to comply with applicable laws, regulations and guidance, Takeda will, at a minimum register all interventional clinical studys it Sponsors anywhere in the world on ClinicalTrials.gov and/or other publicly accessible websites before start of study, as defined in Takeda Policy/Standard. Takeda contact information, along with investigator's city, state (for American investigators), country, and recruiting status will be registered and available for public viewing.

For some registries, Takeda will assist callers in locating study sites closest to their homes by providing the investigator name, address, and phone number to the callers requesting study information. Once subjects receive investigator contact information, they may call the site requesting enrollment into the study. The investigative sites are encouraged to handle the study inquiries according to their established subject screening process. If the caller asks additional questions beyond the topic of study enrollment, they should be referred to the Sponsor.

Any investigator who objects to the Sponsor providing this information to callers must provide the Sponsor with a written notice requesting that their information not be listed on the registry site.

### 13.4.3 Clinical Trial Results Disclosure

Takeda will post the results of clinical studies on ClinicalTrials.gov or other publicly accessible websites, as required by Takeda Policy/Standard, applicable laws and/or regulations.

### 13.5 Insurance and Compensation for Injury

Refer to the study site agreement regarding the Sponsor's policy on subject compensation and treatment for injury. If the investigator has questions regarding this policy, he or she should contact the Sponsor or Sponsor's designed.

### ADMINISTRATIVE AND REFERENCE INFORMATION 14.0

### 14.1 **Administrative Information**

# 14.1.1 Study Contact Information

Property of Takeda. For non-commercial use only and subject to the adopte

I confirm that I have read and that I understand this protocol, the Investigator's Brochure, package insert and any other product information provided by the Sponsor. I agree to conduct this study is accordance with the requirements of this protocol and also to protocol.

- The ethical principles that have their origin in the Declaration of Helsinki.
- International Council for Harmonisation, E6 Good Clinical Practice: Consolidated Guideline.
- All applicable laws and regulations, including, without limitation, data privacy laws and regulations.
- Regulatory requirements for reporting serious adverse events defined in Section 10.2.9 of this protocol.
- Terms outlined in the study site agreement.
- Responsibilities of the Investigator (Appendix A).

I further authorize that my personal information may be processed and transferred in accordance with the uses contemplated in Appendix C of this protocol.

| Signature of Investigator | Date |
|---------------------------------------------|-------------|
| ial in the second | |
| Investigator Name (print or type) | |
| Mille | |
| Investigator's Title | <del></del> |
| 2017.0 | |
| Location of Facility (City, State/Provence) | |
| · Ko. | |
| Location of Facility (Country) | <del></del> |
| 0 | |

The Sponsor will perform all study-related activities with the exception of those identified in the Study-Related Responsibilities template. The vendors identified for specific study-related activities will perform these activities in full or in partnership with the Sponsor.

 and subject to the applic

### 14.1.4 List of Abbreviations

AE Adverse event

**ADL** Activities of Daily Living **ALT** Alanine aminotransferase **ANOVA** Analysis of variance

**AST** Aspartate aminotransferase

**AUC** Area under the concentration-time curve

AUC<sub>%extrap</sub> Percent of  $AUC_{\infty}$  extrapolated

Area under the concentration-time curve, from time 0 to the last observed non-zero  $AUC_{last}$ 

concentration

Area under the concentration-time curve, from time 0 extrapolated to infinity  $AUC_{inf}$ 

**BBB** Blood brain barrier **BMI** Body mass index bpm Beats per minute

**CFR** Code of Federal Regulations

CI Confidence interval

Centimeter cm

and subject Maximum observed concentration  $C_{max}$ 

**CRF** Case report form **CRU** Clinical Research Unit

Common Terminology Criteria for Adverse Events **CTCAE** 

CVIntra-subject variability **ECG** Electrocardiogram

FDA Food and Drug Administration **FSH** Follicle-stimulating hormone

Gram(s) g

GCP Good Clinical Practice Hepatitis B surface antigen **HBsAg** Human chorionic gonadotropin hCG

**HCV** Hepatitis C virus

HIV Human immunodeficiency virus

IBInvestigator's Brochure Informed Consent Form

International Council for Harmonisation

**Independent Ethics Committee** Institutional Review Board

Apparent first-order terminal elimination rate constant

kg

LFT Liver function test(s)

ln Natural log **INR** International normalized ratio

LSM Least-squares  $m^2$ Meters squared

MedDRA® Medical Dictionary for Regulatory Activities®

Milligram mg Milliliter mL

Millimeter of mercury mmHg

msec Millisecond Sample size n NA Not applicable **NMDA** N-methyl-D-aspartate

ΟZ

OATP Organic anion-transporting polypeptide

PK Pharmacokinetic(s) РО Oral administration PPI Proton pump inhibitor PT Prothrombin time QD Once daily

and subject to the applicant QT interval corrected for heart rate using Fridericia's formula QTcF

SAE Serious adverse event Statistical analysis plan SAP

Suspected unexpected serious adverse reactions **SUSAR** Apparent first-order terminal elimination half-life

Treatment-emergent adverse event **TEAE** 

Time to reach maximum observed concentration [C<sub>max</sub>]

gent adv ch maximum Limit of normal United States United States of America World Health Organization

### 15.0 DATA HANDLING AND RECORDKEEPING

The full details of procedures for data handling will be documented in the Data Management Plan.

### 15.1 CRFs (Electronic and/or Paper)

The Sponsor or its designee will supply investigative sites with access to CRFs. The Sponsor or its designee will train appropriate site staff in the use of the CRF. These forms are used to transmit the information collected in the performance of this study to the Sponsor and regulatory authorities. CRFs must be completed in English.

After completion of the entry process, computer logic checks will be run to identify items, such as inconsistent dates, missing data, and questionable values. Queries may be issued by Takeda personnel (or designees) and will be answered by the site.

Corrections are recorded in an audit trail that captures the old information, the new information, identification of the person making the correction, the date the correction was made, and the reason for change. Reasons for significant corrections should additionally be included.

The principal investigator must review the CRFs for completeness and accuracy and must sign and date the appropriate CRFs as indicated. Furthermore, the investigator must retain full responsibility for the accuracy and authenticity of all data entered on the CRFs.

After the lock of the clinical study database, any change of, modification of, or addition to the data on the CRFs should be made by the investigator with use of change and modification records of the CRFs. The principal investigator must review the data change for completeness and accuracy, and must sign and date.

CRFs will be reviewed for completeness and acceptability at the study site during periodic visits by study monitors. The Sponsor of its designee will be permitted to review the subject's medical and hospital records pertinent to the study to ensure accuracy of the CRFs. The completed CRFs are the sole property of the Sponsor and should not be made available in any form to third parties, except for authorized representatives of appropriate governmental health or regulatory authorities, without written permission of the Sponsor.

### 15.2 Record Retention

The investigator agrees to keep the records stipulated in Section 15.1 and those documents that include (but are not limited to) the study-specific documents, the identification log of all participating subjects, medical records, temporary media such as thermal sensitive paper, source worksheets, all original signed and dated informed consent forms, subject authorization forms regarding the use of personal health information (if separate from the informed consent forms), copy of CRFs, including the audit trail, and detailed records of drug disposition to enable evaluations or audits from regulatory authorities, the Sponsor or its designees. Any source documentation printed on degradable thermal sensitive paper should be photocopied by the site and filed with the original in the subject's chart to ensure long-term legibility. Furthermore, ICH E6 Section 4.9.5 requires the investigator to retain essential documents specified in ICH E6 (Section 8) until at least 2 years after the last approval of a marketing application for a specified

Use Investigation is discontinued and regulatory authorities are notified. In addition, ICH E6
Section 4.9.5 states that the study records should be retained until an amount of time specified by applicable regulatory requirements or for a time specified in the Clinical Study Site Agreement between the investigator and Sponsor.

Refer to the Clinical Study Site Agreement

The investigation is not approved, until at least 2 years after une investigation is discontinued and regulatory authorities are notified. In addition, ICH E6
Section 4.9.5 states that the study records should be retained until an amount of time specified by applicable regulatory requirements or for a time specified in the Clinical Study Site Agreement.

The investigation is discontinued and regulatory authorities are notified. In addition, ICH E6
Section 4.9.5 states that the study records should be retained until an amount of time specified by applicable regulatory requirements or for a time specified in the Clinical Study Site Agreement.

 and subject to the appropriate the second seco The investigator and the head of the institution should contact and receive written approval from

### 16.0 REFERENCES

- 1. Parkman HP, Hasler WL, Fisher RS, American Gastroenterological A. American Gastroenterological Association technical review on the diagnosis and treatment of gastroparesis. Gastroenterology 2004;127(5):1592-622.
- 2. Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L, American College of G. Clinical guideline: management of gastroparesis. Am J Gastroenterol 2013;108(1):18-37; quiz 8.
- 3. Hyett B, Martinez FJ, Gill BM, Mehra S, Lembo A, Kelly CP, et al. Delayed radionucleotide gastric emptying studies predict morbidity in diabetics with symptoms of gastroparesis. Gastroenterology 2009;137(2):445-52.
- 4. Takeda Pharmaceuticals, Inc. Global Investigator Brochure. Edition 2.0, July 2018.
- 5. NEXIUM® delayed-release 20 and 40 mg capsules, AstraZeneca Pharms, label, 07 June 2018 Available at: https://www.accessdata.fda.gov/drugsatfda\_docs/label/2018/021153s053,022101s017,02195 7s020lbl.pdf
- 6. NEXIUM® FDA review of NDA 21-153/21-154 for AstraZeneca Pharmaceuticals Esomeprazole Magnesium Delayed-Release Capsules, March 12, 1999. Available at: http://www.accessdata.fda.gov/scripts/cder/drugsatfda/.
- 7. Andersson T1, Röhss K, Bredberg E, Hassan-Alin M. Pharmacokinetics and pharmacodynamics of esomeprazole, the S-isomer of omeprazole. Aliment Pharmacol Ther. 2001 Oct;15(10):1563-9
- 8. Wilder-Smith CH1, Röhss K, Nilsson-Pieschl C, Junghard O, Nyman L. Esomeprazole 40 mg provides improved intragastric acid control as compared with lansoprazole 30 mg and rabeprazole 20 mg in healthy volunteers. Digestion. 2003;68(4):184-8. Epub 2003 Dec 19.
- 9. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 toxicity grading scale. 27Nov2017.

### 17.0 **APPENDICES**

reins of Use

Property of Takeda: For noncommercial use only and subject to the applic

### Appendix A Responsibilities of the Investigator

Clinical research studies sponsored by the Sponsor are subject to ICH GCP and all the applicable local laws and regulations. The responsibilities imposed on investigators by the FDA are summarized in the "Statement of Investigator" (Form FDA 1572), which must be completed and signed before the investigator may participate in this study.

The investigator agrees to assume the following responsibilities by signing a Form FDA 1572:

- 1. Conduct the study in accordance with the protocol.
- 2. Personally conduct or supervise the staff that will assist in the protocol.
- 3. If the investigator/institution retains the services of any individual or party to perform study -related duties and functions, the investigator/institution should ensure that this individual or party is qualified to perform those study -related duties and functions and should implement procedures to ensure the integrity of the study-related duties and functions performed and any data generated.
- 4. Ensure that study related procedures, including study specific (nonroutine/nonstandard panel) screening assessments are NOT performed on potential subjects, prior to the receipt of written approval from relevant governing bodies/authorities.
- 5. Ensure that all colleagues and employees assisting in the conduct of the study are informed of these obligations.
- 6. Secure prior approval of the study and any changes by an appropriate IRB/IEC that conform to 21 CFR Part 56, ICH, and local regulatory requirements.
- 7. Ensure that the IRB/IEC will be responsible for initial review, continuing review, and approval of the protocol. Promptly report to the IRB/IEC all changes in research activity and all anticipated risks to subjects. Make at least yearly reports on the progress of the study to the IRB/IEC, and issue a final report within 3 months of study completion.

Ensure that requirements for informed consent, as outlined in 21 CFR Part 50, ICH and local regulations, are met

- 8. Obtain valid informed consent from each subject who participates in the study, and document the date of consent in the subject's medical chart. Valid informed consent is the most current version approved by the IRB/IEC. Each informed consent form should contain a subject authorization section that describes the uses and disclosures of a subject's personal information (including personal health information) that will take place in connection with the study. If an informed consent form does not include such a subject authorization, then the investigator must obtain a separate subject authorization form from each subject or the subject's legally acceptable representative.
- 9. Prepare and maintain adequate case histories of all persons entered into the study, including CRFs, hospital records, laboratory results, etc, and maintain these data for a minimum of 2 years following notification by the Sponsor that all investigations have been discontinued or that the regulatory authority has approved the marketing application. The investigator should

- 12. P.

  10. Allow possible inspection and copying by the regulatory authority of GCP-specified essential documents.

  11. Maintain current records of the receipt, administration and diagrams, and return all unused Spansor. Properly of Takeda. For non-commercial use only and subject to the appropriate the property of Takeda.
  - 12. Report adverse reactions to the Sponsor promptly. In the event of an SAE, notify the Sponsor

### **Appendix B** Elements of the Subject Informed Consent

In seeking informed consent, the following information shall be provided to each subject, as applicable:

- 1. A statement that the study involves research.
- 2. An explanation of the purposes of the research.
- 4. A description of the procedures to be followed, including invasive procedures.
  5. The identification of any procedures that are
- 6. The estimated number of subjects involved in the study.
- 7. A description of the subject's responsibilities.
- 8. A description of the conduct of the study.
- 9. A statement describing the treatment(s) and the probability for random assignment to each treatment
- 10. A description of the possible side effects of the treatment that the subject may receive.
- 11. A description of any reasonably foreseeable risks or discomforts to the subject and, when applicable, to an embryo, fetus, or nursing infant.
- 12. A description of any benefits to the subject or to others that reasonably may be expected from the research. When there is no intended clinical benefit to the subject, the subject should be made aware of this.
- 13. Disclosures of appropriate alternative procedures or courses of treatment, if any, that might be advantageous to the subject and their important potential risks and benefits.
- 14. A statement describing the extent to which confidentiality of records identifying the subject will be maintained, and a note of the possibility that regulatory agencies, auditor(s), IRB/IEC, and the monitor may inspect the records. By signing a written informed consent form, the subject or the subject's legally acceptable representative is authorizing such access.
- 15. For research involving more than minimal risk, an explanation as to whether any compensation and an explanation as to whether any medical treatments are available if injury occurs and, if so, what they consist of or where further information may be obtained.
- 16. The anticipated prorated payment(s), if any, to the subject for participating in the study.
- 17. The anticipated expenses, if any, to the subject for participating in the study.
- 18. An explanation of whom to contact for answers to pertinent questions about the research (investigator), subject's rights, and IRB/IEC and whom to contact in the event of a research-related injury to the subject.

- 19. A statement that participation is voluntary, that refusal to participate will involve no penalty or loss of benefits to which the subject otherwise is entitled, and that the subject or the subject's legally acceptable representative may discontinue participation at any time without penalty or loss of benefits to which the subject is otherwise entitled.
- 20. The consequences of a subject's decision to withdraw from the research and procedures for orderly termination of participation by the subject.
- 21. A statement that the subject or the subject's legally acceptable representative will be informed in a timely manner if information becomes available that may be relevant to the subject's willingness to continue participation in the study.
- 22. A statement that results of DNA analysis will not be disclosed to an individual, unless prevailing laws require the Sponsor to do so.
- 23. The foreseeable circumstances or reasons under which the subject's participation in the study may be terminated.
- 24. A written subject authorization (either contained within the informed consent form or provided as a separate document) describing to the subject the contemplated and permissible uses and disclosures of the subject's personal information (including personal health information) for purposes of conducting the study. The subject authorization must contain the following statements regarding the uses and disclosures of the subject's personal information:
  - a) that personal information (including personal health information) may be processed by or transferred to other parties in other countries for clinical research and safety reporting purposes, including, without limitation, to the following: (1) Takeda, its affiliates, and licensing partners; (2) business partners assisting Takeda, its affiliates, and licensing partners; (3) regulatory agencies and other health authorities; and (4) IRBs/IECs;
  - b) it is possible that personal information (including personal health information) may be processed and transferred to countries that do not have data protection laws that offer subjects the same level of protection as the data protection laws within this country; however, Takeda will make every effort to keep your personal information confidential, and your name will not be disclosed outside the clinic unless required by law;
  - c) that personal information (including personal health information) may be added to Takeda's research databases for purposes of developing a better understanding of the safety and effectiveness of the study medication(s), studying other therapies for patients, developing a better understanding of disease, and improving the efficiency of future clinical studies;
  - d) that subjects agree not to restrict the use and disclosure of their personal information (including personal health information) upon withdrawal from the study to the extent that the restricted use or disclosure of such information may impact the scientific integrity of the research; and
  - e) that the subject's identity will remain confidential in the event that study results are published.

- Duffeed consent throughout the duration of the study and through to the nonow-up visit (ie, 10-14 days after the last dose of TAK-906).

  26. A statement that clinical study information from this study will be publicly disclosed in a publicly accessible website, such as ClinicalTrials.gov.

 and subject to the applic

### **Appendix C** Investigator Consent to the Use of Personal Information

Takeda will collect and retain personal information of investigator, including his or her name, address, and other personally identifiable information. In addition, investigator's personal information may be transferred to other parties located in countries throughout the world (eg, the United Kingdom, United States, and Japan), including the following:

- Takeda, its affiliates, and licensing partners.
- Business partners assisting Takeda, its affiliates, and licensing partners.
- Regulatory agencies and other health authorities.
- IRBs and IECs.

Investigator's personal information may be retained, processed, and transferred by Takeda and these other parties for research purposes including the following:

- Assessment of the suitability of investigator for the study and/or other clinical studies.
- Management, monitoring, inspection, and audit of the study.
- Analysis, review, and verification of the study results.
- Safety reporting and pharmacovigilance relating to the study.
- Preparation and submission of regulatory filings, correspondence, and communications to regulatory agencies relating to the study.
- Preparation and submission of regulatory filings, correspondence, and communications to regulatory agencies relating to other medications used in other clinical studies that may contain the same chemical compound present in the study medication.
- Inspections and investigations by regulatory authorities relating to the study.
- Self-inspection and internal audit within Takeda, its affiliates, and licensing partners.
- Archiving and audit of study records.
- Posting investigator site contact information, study details and results on publicly accessible clinical study registries, databases, and websites.

Investigator's personal information may be transferred to other countries that do not have data protection laws that offer the same level of protection as data protection laws in investigator's own country.

Investigator acknowledges and consents to the use of his or her personal information by Takeda and other parties for the purposes described above.

# **Appendix D Pregnancy and Contraception Contraception and Pregnancy Avoidance Procedure**

Male Subjects and Their Female Partners

From signing of informed consent, throughout the duration of the study, and through to the follow-up visit, nonsterilized\*\* male subjects who are sexually active with a female partner of childbearing potential\* must use barrier contraception (eg, condom with spermicidal cream or jelly). In addition, they must be advised not to donate sperm during this period. Females of childbearing potential who are partners of male subjects are also advised to use additional contraception as shown in the list containing highly effective/effective contraception below.

Female Subjects and Their Male Partners

- \*A woman is considered a woman of childbearing potential (WOCBP), ie, fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral oophorectomy, hysteroscopic sterilization, and bilateral tubal ligation or bilateral salpingectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range (FSH >40 IU/L) may be used to confirm a post-menopausal state in younger women (eg, those <45 year old) or women who are not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
- \*\* Sterilized males should be at least 1 year post-bilateral vasectomy and have confirmed that they have obtained documentation of the absence of sperm in the ejaculate or have had bilateral orchidectomy.
- 1. Unacceptable methods of contraception are:
  - Spermicides only
  - Withdrawal.
  - No method at all.
  - Use of female and male condoms together.
  - Cap/diaphragm/sponge without spermicide and without condom.
  - Sexual abstinence is NOT an acceptable method of contraception.
- 2. Subjects will be provided with information on highly effective/effective methods of contraception as part of the subject informed consent process and will be asked to sign a consent form stating that they understand the requirements for avoidance of pregnancy, donation of ova, and sperm donation during the course of the study.
- 3. During the course of the study, regular serum human chorionic gonadotropin (hCG) pregnancy tests will be performed for all women only and all subjects (male and female) will receive

reins of Use continued guidance with respect to the avoidance of pregnancy and sperm donation as part of the study procedures. Such guidance should include a reminder of the following:

- a) contraceptive requirements of the study.
- b) reasons for use of barrier methods (ie, condom) in males with pregnant partners.
- c) assessment of subject compliance through questions such as
  - i. Have you used the contraception consistently and correctly since the last visit?
  - ii. Have you forgotten to use contraception since the last visit?
  - iii. Is there a chance for a female partner who could become pregnant?

### **Pregnancy**

Women of childbearing potential will not be included in this study.

Any pregnancies in the partner of a male subject during the study and until the follow up visit, should be recorded following authorization from the subject's partner.

If female partner of a male subject agrees to the primary care physician being informed, the investigator should notify the primary care physician that the subject was participating in a clinical study at the time his female partner became pregnant and provide details of the study drug the subject received (blinded or unblinded, as applicable).

All pregnancies in female partners of male subjects will be followed up to final outcome, using the e birth e birth of Lakeda. For non-commerce property of Lakeda. pregnancy form. The outcome, including any premature termination, must be reported to the sponsor. An evaluation after the birth of the child will also be conducted.

# ELECTRONIC SIGNATURES

| | | ose Pharmacokinetics of Oral TAK-90 | 6 in Healthy Adult Subjects | |
|---|---|---|---|---|
| | | | | SOUSE |
| | | | 25 | 5 |
| | ] | ELECTRONIC SIGNATURES | <0\). | |
| Signed | d by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'UTC') | |
| PPD | | Clinical Pharmacology Approval | 06-Feb-2019 13:58 UTC | |
| | | Clinical Science Approval | 06-Feb-2019 15:31 UTC | |
| Signed PPD | | Biostatistics Approval | 07-Feb-2019 03:03 UTC | |
| | | 1 | *0 | |
| | | .00 | | |
| | | 292 | | |
| | | 31. | | |
| | | Cally . | | |
| | | .00 | | |
| | | ZCjo | | |
| | | Ö | | |
| | con. | | | |
| 4 | , 100 | | | |
| .<0 | )` | | | |
| 99. | | | | |
| , He | | | | |
| ×4 | | | | |
| oel. | | | | |
| OKOK | | | | |